| | Statistical Analysis Flati Fillal |
|---|---|
| <b>gsk</b> GlaxoSmithKline | Statistical Analysis Plan |
| Detailed Title: | A Phase 1/2, randomized, observer-blind, controlled, multi-center study to evaluate safety, reactogenicity and immunogenicity of GSK Biologicals' (RSV) investigational vaccine based on the RSV viral proteins F, N and M2-1 encoded by chimpanzee-derived adenovector (ChAd155-RSV) (GSK3389245A), when administered intramuscularly <i>as</i> a single dose or as two doses according to a 0, 1-month schedule, to infants aged 6 and 7 month |
| eTrack study number and<br>Abbreviated Title | 204894 (RSV PED-011) |
| Scope: | All data pertaining to the above study |
| Date of Statistical Analysis<br>Plan | Final: 27 March 2019 |
| Co-ordinating author: | PPD (Statistician) |
| Reviewed by: | PPD (Clinical and Epidemiology Project Lead); PPD (Clinical Research and Development Lead); PPD (Lead statistician); PPD (Lead statistical analyst); PPD (Scientific writer); PPD (Regulatory Affairs); PPD (SERM physician); PPD - safety scientist; PPD (Public disclosure representative) |
| Approved by: | PPD (Clinical and Epidemiology Project Lead); PPD (Lead statistician); PPD (Study Statistician); PPD (Lead Scientific writer); PPD (Lead statistical Analyst) |

APP 9000058193 Statistical Analysis Plan Template (Effective date: 5th March 2019)

204894 (RSV-PED-011) Statistical Analysis Plan Final

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| LIS | T OF A | BBREVIA | ATIONS | 13 |
| 1. | DOC | JMENT H | ISTORY | 14 |
| 2. | STUD | Y DESIG | N | 14 |
| 3. | OR IE | CTIVES/E | ENDPOINTS | 21 |
| ٥. | 3.1. | _ | /es | |
| | 0.1. | 3.1.1. | Primary Objective | |
| | | 3.1.2. | Secondary Objective | |
| | | 3.1.3. | Tertiary objective | |
| | 3.2. | Endpoin | ıts | |
| | | 3.2.1. | Primary endpoints | |
| | | 3.2.2. | Secondary endpoints | |
| | | 3.2.3. | Tertiary endpoints | 23 |
| 4. | ANAI | YSIS SET | TS | 23 |
| • | 4.1. | | on | |
| | | 4.1.1. | Exposed Set | |
| | | 4.1.2. | Exposed Set of subjects with a negative RSV exposure | |
| | | | status | |
| | | 4.1.3. | Per-protocol Set for analysis of immunogenicity | |
| | 4.2. | | for eliminating data from Analysis Sets | |
| | | 4.2.1. | Elimination from Exposed Set (ES) | 25 |
| | | 4.2.2. | Elimination from Exposed Set (ES) subjects with a | 0.5 |
| | | 400 | negative RSV exposure status | 25 |
| | | 4.2.3. | Elimination from Per-protocol analysis Set (PPS) | 25<br>25 |
| | | | 4.2.3.1. Excluded subjects | 20 |
| 5. | STAT | | ANALYSES | |
| | 5.1. | Demogr | aphy | 27 |
| | | 5.1.1. | Analysis of demographics/baseline characteristics planned | |
| | | | in the protocol | |
| | | 5.1.2. | | |
| | 5.2. | | genicity | |
| | | 5.2.1. | Analysis of immunogenicity planned in the protocol | |
| | | | 5.2.1.1. Within groups assessment | |
| | | | 5.2.1.1.2. Analysis of secondary objectives | |
| | | 5.2.2. | Additional considerations | |
| | 5.3. | - | s of safety and reactogenicity | |
| | 0.0. | 5.3.1. | Analysis of safety and reactogenicity planned in the | |
| | | | protocol | 30 |
| | | | 5.3.1.1. Within groups assessment | 30 |
| | | | 5.3.1.2. Between groups assessment | |
| | | 5.3.2. | Additional considerations | 32 |
| | | | 5.3.2.1. Combined Solicited and Unsolicited Adverse | |
| | | | Events | 33 |

| | | | 5.3.2.2. | Exclusion of implausible solicited Adverse Event | 33 |
|---|---|---|---|---|---|
| | | | 5.3.2.3. | Solicited Adverse Events | |
| | | | 5.3.2.4. | Unsolicited Adverse Events | 34 |
| | 5.4. | Analysis | of RTI and | LRTI | 35 |
| | | 5.4.1. | Analysis o | f RTI and LRTI planned in protocol | 35 |
| | | 5.4.2. | Additional | consideration | 36 |
| 6. | ANAL` | YSIS INTE | ERPRETAT | ION | 36 |
| 7. | COND | | | <b>)</b> | |
| | 7.1. | | | es | |
| | 7.2. | Statistica | al considera | tions for interim analyses | 37 |
| 8. | CHAN | GES FRO | M PLANN | ED ANALYSES | 37 |
| 9. | _ | _ | | ERIVATION RULES AND STATISTICAL | 20 |
| | МЕТН<br>9.1. | | | | |
| | 9.1.<br>9.2. | | | | |
| | 9.2.<br>9.3. | | | ochemistry parameters | |
| | 9.4. | | | f specific interest | |
| 10 | ΔNNE | YES | | | 46 |
| 10. | 10.1. | | | tandard data derivations and statistical methods | |
| | 10.1. | | | events to vaccine doses | |
| | | 10.1.2. | | of missing data | |
| | | | | Dates | |
| | | | 10.1.2.2. | | |
| | | | 10.1.2.3. | Daily recording of solicited symptoms | |
| | | | | 10.1.2.3.1. Studies with paper diaries | |
| | | | 10.1.2.4. | Unsolicited adverse events | |
| | | 10.1.3. | Data deriv | ration | |
| | | | 10.1.3.1. | Age at vaccination in days | 48 |
| | | | 10.1.3.2. | Age at vaccination in months | 48 |
| | | | 10.1.3.3. | Age at vaccination in years | 48 |
| | | | 10.1.3.4. | Weight | |
| | | | 10.1.3.5. | Height | 49 |
| | | | 10.1.3.6. | Body mass index (BMI) | 49 |
| | | | 10.1.3.7. | Temperature | |
| | | | 10.1.3.8. | Numerical serology results | 49 |
| | | | 10.1.3.9. | Geometric mean titers (GMTs) and | |
| | | | | concentrations (GMCs) | |
| | | | | Onset day | |
| | | | | Duration of events | 50 |
| | | | 10.1.3.12. | Counting rules for combining solicited and | |
| | | | | unsolicited adverse events | 50 |
| | | | 10.1.3.13. | Counting rules for occurrences of solicited | |
| | | | | adverse events | |
| | | | | Display of decimals | |
| | | | | Percentages | |
| | | | 10.1.3.16. | Differences in percentages | 51 |

| | ~ · | |
|-----|------------------------------------------------------------|------|
| | 204894 (RSV-PED-0 | |
| | Statistical Analysis Plan F | mai |
| | 10.1.3.17. Demographic/baseline characteristics statistics | |
| | 10.1.3.18. Serological summary statistics | . 52 |
| | 10.1.3.19. Statistical methodology | .52 |
| | 10.1.3.20. Exact confidence intervals around proportions | |
| | 10.1.3.21. Standardized asymptotic confidence intervals | |
| | around differences in proportions | . 52 |
| | 10.2. TFL and/or TFL ToC | |
| 11. | REFERENCES | .54 |
| 12. | LIST OF LISTINGS FOR THE FINAL ANALYSIS | . 55 |
| 12 | MOCK TARLES | 56 |

204894 (RSV-PED-011) Statistical Analysis Plan Final

# **LIST OF TABLES**

| | | PAGE |
|---|---|---|
| Table 1 | Vaccines administered and vaccination schedules | 15 |
| Table 2 | Study groups and epochs foreseen in the study | 16 |
| Table 3 | Study groups and treatment foreseen in the study | 17 |
| Table 4 | Maximum allowed interval between study visits for PPS | 24 |
| Table 5 | Implausible Solicited Adverse Events | 33 |
| Table 6 | Case definitions for data analysis | 38 |
| Table 7 | Toxicity grading scales for hematology and biochemistry parameters applicable for this study | 39 |

204894 (RSV-PED-011) Statistical Analysis Plan Final

# **LIST OF FIGURES**

| | | PAGE |
|----------|--------------|------|
| Figure 1 | Study design | 14 |

204894 (RSV-PED-011) Statistical Analysis Plan Final

# **LIST OF TEMPLATES**

| | | PAGE |
|---|---|---|
| Template 1 | Number of subjects by country and center - <rsv 1d,="" 2d,="" comparator="" placebo="" rsv=""> groups (Exposed Set)</rsv> | 56 |
| Template 2 | Summary of study completion with reasons for withdrawal <rsv 1d,="" 2d,="" comparator="" placebo="" rsv=""> <groups> &lt; pooled RSV 1D, RSV 2D, Comparator/Placebo groups&gt; (Exposed Set)</groups></rsv> | 56 |
| Template 3 | Summary of visit attendance/phone contact completion <rsv 1d,="" 2d,="" comparator="" placebo="" rsv=""> groups (Exposed Set)</rsv> | 57 |
| Template 4 | Summary of important protocol deviations leading to elimination from any analyses <rsv 1d,="" 2d,="" comparator="" placebo="" rsv=""> <groups>&lt; -pooled RSV 1D, RSV 2D, Comparator/Placebo groups&gt;</groups></rsv> | 58 |
| Template 5 | Summary of subject disposition from enrolled set to randomized set (Exposed Set) | 58 |
| Template 6 | Summary of subject disposition from randomized set to exposed set | 59 |
| Template 7 | Summary of subject disposition from Exposed Set to Per<br>Protocol Set at <day 31="" 61="" day="" end="" first="" of="" rsv="" season=""> <rsv<br>1D, RSV 2D, Comparator/Placebo&gt; groups (Exposed set)</rsv<br></day> | 59 |
| Template 8 | Summary of subject disposition from Exposed Set to End of study <rsv 1d,="" 2d,="" comparator="" placebo="" rsv=""> groups (Exposed set)</rsv> | 60 |
| Template 9 | Deviations from protocol for age and intervals between study visits <rsv 1d,="" 2d,="" comparator="" placebo="" rsv=""> groups (Exposed Set)</rsv> | 61 |
| Template 10 | Minimum and maximum visit dates <rsv 1d,="" 2d,="" comparator="" placebo="" rsv=""> groups (Exposed Set)</rsv> | 61 |
| Template 11 | Summary of demographic characteristics - <rsv 1d,="" 2d,="" comparator="" placebo="" rsv=""> <groups>&lt; -pooled RSV 1D, RSV 2D, Comparator/Placebo groups&gt; (Exposed Set, PPS for immunogenicity at <day 31="" 61="" day="" end="" first="" of="" rsv="" season="">)</day></groups></rsv> | 62 |
| Template 12 | Summary of vital signs characteristics - <rsv 1d,="" 2d,="" comparator="" placebo="" rsv=""> <groups>&lt; pooled RSV 1D, RSV 2D, Comparator/Placebo groups&gt; (Exposed set, PPS for immunogenicity at <day 31="" 61="" day="" end="" first="" of="" rsv="" season="">)</day></groups></rsv> | 63 |
| Template 13 | Number of enrolled subjects by age category <rsv 1d,="" 2d,="" comparator="" placebo="" rsv=""> groups</rsv> | 64 |

| Template 14 | Compliance in completing solicited adverse events information <rsv 1d,="" 2d,="" comparator="" placebo="" rsv=""> groups (Exposed Set)64</rsv> |
|---|---|
| Template 15 | Summary of <grade 3=""> adverse events (solicited and unsolicited) <with attend="" causal="" medically="" relationship="" to="" vaccination,="" visit="" with=""> within &lt;7, 30&gt; days following first and second vaccination and overall <rsv 1d,="" 2d,="" comparator="" placebo="" rsv=""> <groups>&lt; pooled RSV 1D, RSV 2D, Comparator/Placebo groups&gt; (Exposed Set)</groups></rsv></with></grade> |
| Template 16 | Percentage of subjects with solicited local adverse events by maximum intensity within the 7-day (Days 1-7) following first and second vaccination and overall - <rsv 1d,="" 2d,="" comparator="" placebo="" rsv=""> <groups> &lt; pooled RSV 1D, RSV 2D, Comparator/Placebo groups&gt;(Exposed Set)</groups></rsv> |
| Template 17 | Duration in days of solicited <general, local=""> adverse events within 7 days following first and second vaccination and overall <rsv 1d,="" 2d,="" comparator="" placebo="" rsv=""> groups (Exposed Set)67</rsv></general,> |
| Template 18 | Percentage of subjects with solicited general adverse events by maximum intensity within the 7-day (Days 1-7) following first and second vaccination and overall - <rsv 1d,="" 2d,="" comparator="" placebo="" rsv=""> <groups> &lt; pooled RSV 1D, RSV 2D, Comparator/Placebo groups &gt;(Exposed Set)</groups></rsv> |
| Template 19 | Percentage of subjects reporting solicited local adverse events (any grade /grade 2,3/ grade 3) within 7-days following first and second vaccination by maximum intensity for pooled RSV 1D, RSV 2D, Comparator/Placebo groups (Exposed Set) |
| Template 20 | Percentage of subjects reporting fever (any and grade 3) and other solicited general adverse events (any grade /grade 2,3/ grade 3) within 7-days following first and second vaccination by maximum intensity for pooled RSV 1D, RSV 2D and Comparator/Placebo groups (Exposed Set) |
| Template 21 | Summary of subjects with at least one <Ø/grade 3/ related/<br>grade 3 related/serious/ medically attended> unsolicited adverse<br>event <episode bleeding="" excessive="" of="" or="" spontaneous=""> classified<br/>by MedDRA Primary System Organ Class and Preferred Term<br/><with 30="" and="" days="" first="" of="" onset="" second="" vaccination="" within=""><from<br>vaccination dose 1 up to Day 61&gt; <pooled> <rsv 1d,="" 2d,<br="" rsv="">Comparator/Placebo&gt; groups (Exposed Set)</rsv></pooled></from<br></with></episode> |
| Template 22 | Summary of subjects with at least one <episode (ae="" adverse="" event="" interest)="" of="" rsv-lrti="" serious="" specific=""> classified by MedDRA Primary System Organ Class and Preferred Term <from 1="" <first="" dose="" end="" of="" second="" to="" up="" vaccination=""> RSV season for pooled RSV 1D, RSV 2D and Comparator/Placebo groups (Exposed Set)</from></episode> |

| Template 23 | Listing of SAE from vaccination dose 1 up to <day 61="" end="" first="" of="" rsv="" season="" study=""> (Exposed Set)</day> | 73 |
|---|---|---|
| Template 24 | Listing of AEs related to LRTI and association to RSV infection from vaccination dose 1 up to <day 61="" end="" first="" of="" rsv="" season="" study=""> (Exposed Set)</day> | 73 |
| Template 25 | Listing of AEs related to spontaneous or excessive bleeding together with hemoglobin and platelet count results with 30 days of first and second vaccination (Exposed Set) | 74 |
| Template 26 | Listing of adverse events, SAEs and solicited symptoms leading to study or treatment discontinuation from vaccination dose 1 up to <day 61="" end="" first="" of="" rsv="" season="" second="">(Exposed Set)</day> | 74 |
| Template 27 | Listing of unscheduled safety visit from vaccination dose 1 up to <day 61="" end="" first="" of="" rsv="" season="" study=""> (Exposed Set)</day> | 74 |
| Template 28 | Summary of subjects taking a concomitant medication within <7/30> days following each vaccination and overall <rsv 1d,="" 2d,="" comparator="" placebo="" rsv=""> <groups>&lt; for pooled RSV 1D, RSV 2D and Comparator/Placebo groups&gt; (Exposed Set)</groups></rsv> | 75 |
| Template 29 | Summary of occurrences and subjects with at least one solicited and unsolicited adverse event classified by MedDRA Primary System Organ Class and Preferred Term with onset within 30 days of first and second vaccination – SAE excluded <rsv 1d,="" 2d,="" comparator="" placebo="" rsv=""> groups (Exposed Set)</rsv> | 76 |
| Template 30 | Number (%) of subjects with serious adverse events <from 1="" 61="" <day="" day="" end="" of="" rsv="" season="" second="" to="" up="">, including number of events reported for pooled RSV 1D, RSV 2D and Comparator/Placebo&gt; groups (Exposed Set)</from> | 77 |
| Template 31 | Number and percentage of subjects with <anti-rsv a="" anti-rsv="" antibody="" concentration="" f="" titre,=""> equal to or above <cut-off><unit> and gm<t,c> for pooled RSV 1D, RSV 2D and Comparator/Placebo&gt; groups (<adapted>PPS of immunogenicity at <day 1st="" end="" of="" rsv="" season="" x,="">)</day></adapted></t,c></unit></cut-off></anti-rsv> | 77 |
| Template 32 | Distribution of <rsv-a antibody="" concentration="" neutralising="" rsv-f="" titre,=""> for pooled RSV 1D, RSV 2D and Comparator/Placebo&gt; groups (<adapted>PPS for immunogenicity <at 1st="" day="" end="" of="" rsv="" season="" x,="">)</at></adapted></rsv-a> | 78 |
| Template 33 | Vaccine response for anti-RSV-A neutralising antibody titre at each post-vaccination timepoint for pooled RSV 1D, RSV 2D and Comparator/Placebo> groups (PPS for analysis of immunogenicity at <day 1st="" end="" of="" rsv="" season="" x,="">)</day> | 79 |
| Template 34 | Number and percentage of subjects with <anti-rsv a="" anti-rsv="" antibody="" concentration="" f="" titre,=""> equal to or above <cut-off< td=""><td></td></cut-off<></anti-rsv> | |

| | > <unit> and GMR for pooled RSV 1D, RSV 2D and Comparator/Placebo&gt; groups (PPS of immunogenicity at <day 1st="" end="" of="" rsv="" season="" x,="">)</day></unit> | 80 |
|---|---|---|
| Template 35 | Distribution of fold of anti-RSV-A neutralising antibody titer by <cumulative> pre-vaccination titer category for pooled RSV 1D, RSV 2D and Comparator/Placebo&gt; groups (PPS for analysis of immunogenicity at <day end="" first="" of="" rsv="" season="" x,="">)</day></cumulative> | 81 |
| Template 36 | Descriptive statistics of <anti-rsv a="" anti-rsv="" antibody="" concentration="" f="" neutralizing="" titre,="">at pre-vaccination, Day &lt;31, 61,&gt; <and 1st="" end="" of="" rsv="" season="" transmission=""> for pooled RSV 1D, RSV 2D and Comparator/Placebo&gt; groups (<adapted> PPS for immunogenicity)</adapted></and></anti-rsv> | 82 |
| Template 37 | Reverse cumulative distribution curves for anti-RSV-A neutralising antibody titres in each group at baseline and <day 31,="" 61,="" day="" end="" first="" of="" rsv="" season=""> for pooled RSV 1D, RSV 2D and Comparator/Placebo&gt; group <pps 1st="" <day="" analysis="" at="" end="" for="" immunogenicity="" of="" rsv="" season="" x,=""></pps></day> | 83 |
| Template 38 | Individual results of anti-RSV-A neutralising antibody titre at Day <61/end of first RSV season> versus pre-vaccination in <each 1d,="" 2d="" <rsv="" pooled="" rsv=""> group&gt; and Comparator/placebo group&gt; (PPS for analysis of immunogenicity at <day x="">)</day></each> | 83 |
| Template 39 | Number and percentage of subjects with at least one RSV infection, RSV-RTI, RSV-LRTI, RSV-severe LRTI, RSV-very severe LRTI, All-cause LRTI and RSV hospitalization (based on WHO case definition) from vaccination dose 1 up to end of <first, second=""> RSV season for pooled RSV 1D, RSV 2D and Comparator/Placebo group (<exposed a="" exposed="" exposure="" negative="" rsv="" set="" set,="" status="" with="">)</exposed></first,> | 84 |
| Template 40 | Proportion of subjects with at least one RSV hospitalization over the number of subjects with at least one RSV infection (symptomatic or asymptomatic*) from vaccination dose 1 up to end of <first, second=""> RSV season for pooled RSV 1D, RSV 2D and Comparator/Placebo group <exposed baseline="" exposed="" negative="" rsv="" set="" set,="" status="" with=""></exposed></first,> | 84 |
| Template 41 | Number and percentage of subjects reporting the RSV infection of different severity (based on WHO case definition) by number of events experienced between vaccination dose 1 up to end of <first, second=""> RSV season for pooled RSV 1D, RSV 2D and Comparator/Placebo group <exposed baseline="" exposed="" negative="" rsv="" set="" set,="" status="" with=""></exposed></first,> | 85 |
| Template 42 | Number and percentage of RSV infections and associated disease severity (based on WHO case definition) and relative risk from vaccination dose 1 up to end of <first, second=""> RSV season for pooled RSV 1D, RSV 2D and Comparator/Placebo</first,> | |

| | group <exposed baseline="" exposed="" negative="" rsv="" set="" set,="" status="" with=""></exposed> | 86 |
|---|---|---|
| Template 43 | Number and percentage of RSV infections (based on WHO case definition) requiring hospitalization between vaccination dose 1 up to end of <first, second=""> RSV season for pooled RSV 1D, RSV 2D and Comparator/Placebo group <exposed baseline="" exposed="" negative="" rsv="" set="" set,="" status="" with=""></exposed></first,> | 86 |
| Template 44 | Descriptive statistics of viral load calculated on all qRT-PCR confirmed RSV infection episodes with varying disease severity (based on WHO case definition) from vaccination dose 1 up to end of <first, second=""> RSV season for pooled RSV 1D, RSV 2D and Comparator/Placebo group <exposed baseline="" exposed="" negative="" rsv="" set="" set,="" status="" with=""></exposed></first,> | 87 |
| Template 45 | Descriptive statistics of maximum viral load per subjects based on qRT-PCR confirmed episode with varying disease severity (based on WHO case definition) form vaccination dose 1 up to end of <first, second=""> RSV season for pooled RSV 1D, RSV 2D and Comparator/Placebo group <exposed baseline="" exposed="" negative="" rsv="" set="" set,="" status="" with=""></exposed></first,> | 88 |
| Template 46 | Frequency of multiple respiratory pathogen for qRT-PCR confirmed RSV-RTI episodes from vaccination dose 1 up to end of <first, second=""> RSV season for pooled RSV 1D, RSV 2D and Comparator/Placebo groups <exposed baseline="" exposed="" negative="" rsv="" set="" set,="" status="" with=""></exposed></first,> | 89 |
| Template 47 | Frequency of multiple respiratory pathogen for confirmed LRTI episodes from vaccination dose 1 up to end of <first, second=""> RSV season for pooled RSV 1D, RSV 2D and Comparator/Placebo groups <exposed baseline="" exposed="" negative="" rsv="" set="" set,="" status="" with=""></exposed></first,> | 90 |
| Template 48 | Listing of RSV-RTI cases identified according to WHO case definitions from vaccination dose 1 up to end of second RSV season <exposed baseline="" exposed="" negative="" rsv="" set="" set,="" status="" with=""></exposed> | 90 |
| Template 49 | Listing of RSV-RTI requiring hospitalization and type of inpatient facility required from vaccination dose 1 up to end of second RSV season <exposed baseline="" exposed="" negative="" rsv="" set="" set,="" status="" with=""></exposed> | 91 |
| Template 50 | Number and percentage of subjects with highest associated severity of RSV infection (based on WHO case definition) from vaccination dose 1 up to <first, second=""> RSV season for pooled RSV 1D, RSV 2D and Comparator/Placebo groups <exposed baseline="" exposed="" negative="" rsv="" set="" set,="" status="" with=""></exposed></first,> | 91 |
| Template 51 | Number and percentage of subjects reporting the RSV infection of maximum severity (based on WHO case definition) by number | |

| | of events experienced between vaccination dose 1 up to end of <first, second=""> RSV season for pooled RSV 1D, RSV 2D and Comparator/Placebo groups <exposed baseline="" exposed="" negative="" rsv="" set="" set,="" status="" with=""></exposed></first,> | . 92 |
|---|---|---|
| Template 52 | Number and percentage of subjects with <anti-rsv a="" anti-rsv="" antibody="" concentration="" f="" titre,=""> equal to or above <cut-off><unit> and gm<t,c> for pooled RSV 1D, RSV 2D and Comparator/Placebo&gt; groups – by RSV baseline status (<adapted>PPS of immunogenicity at <day 1st="" end="" of="" rsv="" season="" x,="">)</day></adapted></t,c></unit></cut-off></anti-rsv> | . 93 |
| Template 53 | Distribution of <rsv-a antibody="" concentration="" neutralising="" rsv-f="" titre,=""> for pooled RSV 1D, RSV 2D and Comparator/Placebo&gt; groups – by RSV baseline status(<adapted>PPS for immunogenicity <at 1st="" day="" end="" of="" rsv="" season="" x,="">)</at></adapted></rsv-a> | . 94 |
| Template 54 | Number and percentage of subjects with <anti-rsv a="" anti-rsv="" antibody="" concentration="" f="" titre,=""> equal to or above <cut-off><unit> and GMR for pooled RSV 1D, RSV 2D and Comparator/Placebo&gt; groups – by RSV baseline status (PPS of immunogenicity at <day 1st="" end="" of="" rsv="" season="" x,="">)</day></unit></cut-off></anti-rsv> | . 95 |
| Template 55 | Descriptive statistics of <anti-rsv a="" anti-rsv="" antibody="" concentration="" f="" neutralizing="" titre,="">at pre-vaccination, Day &lt;31, 61,&gt; <and 1<sup="" end="" of="">st RSV transmission season&gt; for pooled RSV 1D, RSV 2D and Comparator/Placebo&gt; groups – by RSV baseline status (<adapted> PPS for immunogenicity)</adapted></and></anti-rsv> | . 96 |
| Template 56 | Summary of subjects by unsolicited adverse event category with onset within 30 days of first and second vaccination (Exposed Set) | .96 |
| Template 57 | Number and percentage of subjects with at least one RSV-RTI progressing to RSV-LRTI, RSV-severe LRTI, RSV-very severe LRTI and RSV hospitalization from vaccination dose 1 up to end of <first, second=""> RSV season for pooled RSV 1D, RSV 2D and Comparator/Placebo groups <es, exposed="" exposure="" negative="" rsv="" set="" status="" with=""></es,></first,> | .97 |

204894 (RSV-PED-011) Statistical Analysis Plan Final

### **LIST OF ABBREVIATIONS**

**AE** Adverse event

**AESI** Adverse Events of Special Interest

**ChAd155-** Investigational recombinant chimpanzee adenovirus Type 155-

**RSV** vectored RSV vaccine

**CI** Confidence Interval

**ERD** Enhanced Respiratory Disease

**ES** Exposed Set

**GMC** Geometric mean antibody concentration

**GMT** Geometric mean antibody titre

**GSK** GlaxoSmithKline

**LL** Lower Limit of the confidence interval

**LLOO** Lower Limit of Quantification

**LRTI** Lower respiratory tract infection

**MedDRA** Medical Dictionary for Regulatory Activities

NA Not Applicable

**PD** Protocol Deviation

**PPS** Per-Protocol Set

**RR** Relative Risk

**RSV** Respiratory Syncytial Virus

**RTI** Respiratory Tract Infection

**SAE** Serious adverse event

**SAP** Statistical Analysis Plan

**SD** Standard Deviation

**SDTM** Study Data Tabulation Model

**SPM** Study Procedure Manual

**SR** Study Report

**TFL** Tables Figures and Listings

**ToC** Table of Content

UL Upper Limit of the confidence interval

**ULOQ** Upper Limit of Quantification

### 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|-------------|-------------|--------------------------|
| 27 MAR 2019 | Final | Amendment 3: 21 MAR 2019 |

### 2. STUDY DESIGN

### Figure 1 Study design



- **D**: Day; **FU**: follow-up; **IDMC**: Independent Data Monitoring Committee; **iSRC**: internal Safety Review Committee; **RSV**: respiratory syncytial virus; **RTI**: respiratory tract infection; **SE**: solicited events; **V**: Visit **1D**: 1 Dose (1.5x10<sup>10</sup> vp/dose); **2D**: 2 Dose (5x10<sup>10</sup> vp/dose); FB: Formulation buffer S9b.
- \* Vaccine Dose 1 at Day 1 will be administered before the first RSV season (refer to Section 5.1 of the protocol for definition of RSV season).
- † Visit 2 (Day 8), Visit 4 (Day 38), and Visit 8 (no blood sampling for immune response and no vaccine administration) may take place in the subject's home or at the investigators clinical facility as appropriate to the circumstances in the judgment of the investigator. For authorized sites only, Visit 5 (Day 61) and Visit 7 (both with blood sampling) may also take place in the subject's home or at the investigators clinical facility as appropriate to the circumstances in the judgment of the investigator
- ‡ In countries where *Menveo* or Placebo is used as a comparator, no administration will be performed at Day 121 and therefore in those countries there will be no Visit 6 and it will be administered at the end of the first RSV season at Visit 7 (refer to Table 2 and Table 7 of the protocol).
- <sup>a</sup> Surveillance for RSV-RTI comprises monthly nasal swab collected to detect asymptomatic RSV infections during RSV season and active and passive surveillance contacts for RSV symptomatic RTI. Of note the swab may be omitted if a nasal swab has been taken at a symptomatic visit in the same month (see Section 9.2 of the protocol). Data about RSV–RTI incidence will be reviewed monthly by an IDMC.
- <sup>b</sup> An iSRC will review all accumulating safety data monthly until the IDMC reviews has reviewed all safety data up to 30 days after administration of Dose 2 (i.e., Day 61). The IDMC will review all accumulating safety data monthly throughout the period of vaccination and accumulating SAEs until the end of the second RSV transmission season. Refer to Sections 9.10.2 and 9.10.3 of the protocol.
- c Refer to Section 6.6.12.3 of the protocol

Table 1 Vaccines administered and vaccination schedules

| 0 | | Age* (Months) / (Visit, Day) | | | |
|---|---|---|---|---|---|
| Groups | 6-7 / (V1, D1) | 7-8 / (V3, D31) | 8-9 / (V5, D61) | 10-11 / (V6, D121)** | 14-18 / (V7) |
| 1D RSV + Bexsero | 1D RSV ChAd | FB | Bexsero | Bexsero | Bexsero |
| 2D RSV + Bexsero | 2D RSV ChAd | 2D RSV ChAd | Bexsero | Bexsero | Bexsero |
| Bexsero | Bexsero | FB | Bexsero | FB | Bexsero |
| 1D RSV + Nimenrix | 1D RSV ChAd | FB | Nimenrix | Nimenrix | Nimenrix |
| 2D RSV + Nimenrix | 2D RSV ChAd | 2D RSV ChAd | Nimenrix | Nimenrix | Nimenrix |
| Nimenrix | Nimenrix | FB | Nimenrix | FB | Nimenrix |
| 1D RSV + Synflorix | 1D RSV ChAd | FB | Synflorix | Synflorix | Synflorix |
| 2D RSV + Synflorix | 2D RSV ChAd | 2D RSV ChAd | Synflorix | Synflorix | Synflorix |
| Synflorix | FB | Synflorix | Synflorix | FB | Synflorix |
| 1D RSV + Menveo | 1D RSV ChAd | FB | Menveo | | Menveo |
| 2D RSV + Menveo | 2D RSV ChAd | 2D RSV ChAd | Menveo | | Menveo |
| Menveo | FB | Menveo | FB | | Menveo |
| 1D RSV + Placebo | 1D RSV ChAd | FB | | | |
| 2D RSV + Placebo | 2D RSV ChAd | 2D RSV ChAd | | | |
| Placebo | FB | FB | | | |

V: Visit; D: Day; 1D: 1 Dose (1.5x10<sup>10</sup> vp/dose); 2D: 2 Dose (5x10<sup>10</sup> vp/dose); RSV ChAd: ChAd155-RSV vaccine; FB: Formulation buffer S9b.

- Experimental design: Phase I/II, observer-blind, randomized, controlled, multicentric study with three parallel groups
- Duration of the study: approximately 24 months.
  - Epoch 001: Screening Visit starting up to 30 days before first vaccination and ending on Day -1.
  - Epoch 002: primary starting at Visit 1 (Day 1) and ending at Visit 5 (Day 61).
  - Epoch 003: follow-up starting after Visit 5 (Day 61)\* and ending at Visit 7 (end of the first RSV transmission season).
  - Epoch 004: follow-up starting after Visit 7 (end of the first RSV transmission season)\* and ending at Visit 8 (end of the second RSV transmission season).
  - \*Any safety, immunogenicity and disease surveillance data collected beyond Visit 5 (Day 61) will be collected in Epoch 003. Any safety, immunogenicity and disease surveillance data collected beyond Visit 7 (end of the first RSV transmission season) will be collected in Epoch 004. Refer to the SPM for RSV transmission seasons per country.
- Primary Completion Date (PCD): Visit 5 (Day 61).

<sup>\*</sup> Assumes enrolled at 6 and 7 months of age for the vaccine Dose 1 to be administered before the first RSV season; the second dose will be given one month after the first dose. (RSV seasons will be determined for each country based on local epidemiological data [The RSV season is defined as the period of the year when 70% of the RSV cases have occurred in previous years. For the calculation, where available, data from up to the ten previous years should be applied. If the data permit calculation of the actual date of the beginning of the season, rather than approximation to the nearest month, this is desirable. Refer to the SPM for RSV seasons per country.])

<sup>\*\*</sup> In countries where *Menveo* or Placebo is used as a comparator, no administration will be performed at Day 121 and therefore in those countries there will be no Visit 6 and it will be administered at the end of the first RSV season at Visit 7.

- End of Study (EoS): Last testing results released of samples collected at Visit 8 (end of the second RSV transmission season) related to primary and secondary endpoints.\*
  - \* Up to Visit 8 (end of the second RSV season), there will be monthly nasal swab to detect asymptomatic RSV infections during the RSV season *or* if following active or a passive surveillance contacts, a subject presents symptoms of respiratory tract infection (RTI), a nasal swab will be collected.
- Study groups:

Table 2 Study groups and epochs foreseen in the study

| Ctudu anauma | Target Number | A are (Min/Mess) | Epochs | | | |
|---|---|---|---|---|---|---|
| Study groups | of subjects | Age (Min/Max) | Epoch 001 | Epoch 002 | Epoch 003 | Epoch 004 |
| 1D RSV + Bexsero | | 6 – 7 months | N/A | Х | Х | Х |
| 1D RSV + Nimenrix | | 6 – 7 months | N/A | Х | Х | х |
| 1D RSV + Synflorix | 50 | 6 – 7 months | N/A | Х | Х | х |
| 1D RSV + Menveo | | 6 – 7 months | N/A | Х | Х | х |
| 1D RSV + Placebo | | 6 – 7 months | N/A | Х | Х | Х |
| 2D RSV + Bexsero | | 6 – 7 months | N/A | Х | Х | Х |
| 2D RSV + Nimenrix | | 6 – 7 months | N/A | Х | Х | х |
| 2D RSV + Synflorix | 50 | 6 – 7 months | N/A | Х | Х | х |
| 2D RSV + Menveo | | 6 – 7 months | N/A | Х | Х | х |
| 2D RSV + Placebo | | 6–7 months | N/A | Х | Х | Х |
| Bexsero | | 6 – 7 months | N/A | Х | Х | Х |
| Nimenrix | | 6 – 7 months | N/A | Х | Х | Х |
| Synflorix | ynflorix 50 | | N/A | Х | Х | Х |
| Menveo | | 6 – 7 months | N/A | Х | Х | Х |
| Placebo | | 6 – 7 months | N/A | Х | Х | Х |

<sup>1</sup>D: 1 Dose (1.5x10<sup>10</sup> vp/dose); RSV: ChAd155-RSV vaccine; 2D: 2 Dose (5x10<sup>10</sup> vp/dose); N/A: Not Applicable.

| Table 3 | Study groups and treatment foreseen in the study |
|---------|--------------------------------------------------|
|---------|--------------------------------------------------|

| Treatment name | 1D RSV ChAd | 2D RSV ChAd | Bexsero | Nimenrix | Synflorix | Menveo | FB |
|---|---|---|---|---|---|---|---|
| | 1D ChAd155-RSV<br>1.5X10 <sup>10</sup> vp/dose | 2D ChAd155-RSV<br>5X10 <sup>10</sup> vp/dose | Bexsero | Nimenrix | Synflorix | Menveo | FB |
| Study Groups | | | | | | | |
| 1D RSV + Bexsero | Х | | X | | | | X |
| 1D RSV + Nimenrix | х | | | х | | | X |
| 1D RSV + Synflorix | х | | | | X | | X |
| 1D RSV + Menveo | х | | | | | X | X |
| 1D RSV + Placebo | х | | | | | | X |
| 2D RSV + Bexsero | | Х | Х | | | | |
| 2D RSV + Nimenrix | | Х | | х | | | |
| 2D RSV + Synflorix | | Х | | | Х | | |
| 2D RSV + Menveo | | х | | | | X | |
| 2D RSV + Placebo | | х | | | | | |
| Bexsero | | | Х | | | | Х |
| Nimenrix | | | | Х | | | X |
| Synflorix | | | | | X | | X |
| Menveo | | | | | | Х | X |
| Placebo | | | | | | | X |

**ChAd155-RSV**: Chimpanzee Adenovirus Type 155 RSV vaccine; **FB**: Formulation buffer S9b; **RSV ChAd**: ChAd155-RSV vaccine; **1D**: 1 Dose (1.5x10<sup>10</sup> vp/dose); **2D**: 2 Dose (5x10<sup>10</sup> vp/dose).

- Controls: active comparator vaccines (*Bexsero*, or *Nimenrix*, or *Synflorix*, or *Menveo*, or Placebo (FB)\*.
  - \* The choice of active comparator vaccine (*Bexsero*, *Nimenrix*, *Synflorix*, or *Menveo*) or Placebo is done at the country level. Refer to the ICF for the local choice of comparator/Placebo.

### Vaccination schedules:

- **RSV investigational vaccine:** In the 1 Dose (1D) groups, a single lower dose of 1.5x10<sup>10</sup> vp will be administered IM at Day 1 (Visit 1). Formulation buffer will be administered in the 1D groups at Day 31 (Visit 3). In the 2 Dose (2D) groups, two doses of 5x10<sup>10</sup> vp will be administered IM according to a 0, 1-month schedule, (i.e., at Day 1 [Visit 1] and Day 31 [Visit 3]) (see Figure 1 and Table 1). Dose 1 will be administered before the first RSV season and the second dose will be given one month after the first dose (RSV seasons will be determined for each country based on local epidemiological data and documented in the Study Procedures Manual [SPM]. The RSV season is defined as the period of the year when 70% of the RSV cases have occurred in previous years. For the calculation, where available, data from up to the ten previous years should be applied. If the data permit calculation of the actual date of the beginning of the season, rather than approximation to the nearest month, this is desirable.)
- Comparator or Placebo: In countries where Bexsero or Nimenrix is used as a control, two doses will be administered IM with at least a 2-month interval between these primary doses. A booster dose will be administered IM in the second year of life at Visit 7, with an interval of at least 2 months between the

204894 (RSV-PED-011) Statistical Analysis Plan Final

primary series and booster dose. The first *Bexsero* or *Nimenrix* dose will be administered at Day 1 (Visit 1) (in the groups receiving only *Bexsero* or *Nimenrix*, respectively). In the groups receiving only *Bexsero* or *Nimenrix*, the second dose will be at Day 61 (Visit 5). The first *Bexsero* or *Nimenrix* dose to be administered to the 1D and 2D RSV groups will be at Day 61 (Visit 5), following the 1 or 2 RSV vaccine doses, respectively. The second dose of *Bexsero* or *Nimenrix* in the 1D and 2D groups will be at Day 121 (Visit 6). Formulation buffer will be administered, when neither RSV vaccine nor comparator is scheduled, at the 5 vaccination visits (see Figure 1 and Table 1).

- In countries where *Synflorix* is used as a control, two doses will be administered IM with at least a 1 month interval between these primary doses. A booster dose will be administered IM in the second year of life at Visit 7. The first *Synflorix* dose will be administered at Day 31 (Visit 3) (in the group receiving only *Synflorix*). In the group receiving only *Synflorix*, the second dose will be at Day 61 (Visit 5). The first *Synflorix* dose to be administered to the 1D and 2D RSV groups will be at Day 61 (Visit 5), following the 1 or 2 RSV vaccine doses, respectively. The second dose of *Synflorix* in the 1D and 2D groups will be at Day 121 (Visit 6). Formulation buffer will be administered, when neither RSV vaccine nor comparator is scheduled, at the 5 vaccination visits (see Figure 1 and Table 1).
- In countries where *Menveo* is used as a control, two doses will be administered IM at least 3 months apart with the second dose in the second year of life at Visit 7. The first *Menveo* dose will be administered at Day 31 (Visit 3) (in the group receiving only *Menveo*). The first *Menveo* dose to be administered to the 1D and 2D RSV groups will be at Day 61 (Visit 5), following the 1 or 2 RSV vaccine doses, respectively. Since the second *Menveo* dose has to be administered in the second year of life at Visit 7, no administration will be performed at Day 121 (Visit 6). Formulation buffer will be administered, when neither RSV vaccine or comparator is scheduled, at the 4 vaccination visits (see Figure 1 and Table 1).
- In countries where Placebo is used as a control, one dose will be administered IM at Day 31 (Visit 3) in the 1D RSV + Placebo group and two IM doses will be administered IM according to a 0, 1-month schedule at Day 1 (Visit 1) and Day 31 (Visit 3) in the Placebo group (see Figure 1 and Table 1).
- Treatment allocation: infants will be randomized using a centralized randomization system on internet (SBIR) before first vaccination and after assessment of eligibility (i.e., after screening conclusion) (refer to Section 6.2.2 of the protocol for details about randomization of treatment). The randomization algorithm will use a minimization procedure accounting for country as a minimization factor and the grouping comparator/placebo as a stratification factor.
- Blinding: not applicable for Epoch 001 (Screening Visit), observer-blind in Epoch 002 and single-blind in Epoch 003 and Epoch 004. Refer to Section 6.3 of the protocol for details of blinding procedure.

## Blinding of study epochs

| Study Epochs | Blinding |
|--------------|----------------|
| Epoch 001 | N/A |
| Epoch 002 | observer-blind |
| Epoch 003 | single-blind |
| Epoch 004 | single-blind |

### Sampling schedule:

- Blood samples for hematology/biochemistry will be taken from all infants at Screening (up to 30 days before first vaccination to Day -1). Blood samples for hematology/biochemistry may be taken from infants at any timepoints, if deemed necessary by the investigator. Refer to Table 12 of the protocol for the list of parameters to be tested.
- Refer to Section 6.6.1.2.2 and Figure 2 of the protocol for information about the re-testing of samples in case of any Grade 1 abnormality with potential clinical relevance (according to investigators judgment) or any ≥ Grade 2 abnormality.
- Blood samples for humoral immunogenicity will be taken from all subjects at Screening and on Day 31, Day 61, and at the visit occurring at the end of the first RSV transmission season.
- Blood sample for assessment of mechanism of illness (potential ERD) will be taken from subjects hospitalized for LRTI (only for RSV-positive subjects using a locally available RSV test).
- Nasal swab: there will be monthly nasal swab to detect asymptomatic RSV infections during the RSV season and if following active or a passive surveillance contacts, a subject present symptoms of RTI, a nasal swab will be collected (as well as a sample for local testing i.e., the type of sample to be determined locally [e.g., swab, etc.]) (Refer to the SPM).
- Study visits: Other than the screening visit and assessment visits for active/passive surveillance, there will be 8 study visits except in countries where *Menveo* or Placebo is used as a control where there will be 7 study visits.
  - In countries where *Menveo* is used as a comparator, no administration will be performed at Day 121 and therefore in those countries there will be no Visit 6 and it will be administered at the end of the first RSV season at Visit 7 (refer to Table 2 and 7 of the protocol).
  - In countries where Placebo is used as a control, no vaccine administration will be performed after Visit 3 and therefore in those countries there will be no Visit 6. There will be a Visit 5 and Visit 7 for countries using Placebo and all other study procedures will occur at these visits except vaccination.
  - Visit 2 (Day 8), Visit 4 (Day 38), and Visit 8 (no blood sampling for immune response and no vaccine administration) may take place in the subject's home or at the investigators clinical facility as appropriate to the circumstances in the judgment of the investigator.

204894 (RSV-PED-011) Statistical Analysis Plan Final

- o For authorized sites only, Visit 5 (Day 61) and Visit 7 (both with blood sampling) may also take place in the subject's home or at the investigators clinical facility as appropriate to the circumstances in the judgment of the investigator.
- o Data collection: electronic Case Report Form (eCRF).
- Safety monitoring: internal safety review committee (iSRC) and IDMC (refer to Section 9.10 of the protocol).
- Surveillance for RSV-RTI, difficulty in breathing, and wheezing episodes
  Surveillance period will be carried out from Visit 1 (after Dose 1) until the last study
  visit (end of the second RSV transmission season). In order to detect asymptomatic
  RSV-RTI, monthly nasal swabs for analysis at sponsor laboratory will be performed
  for all subjects during the RSV season. In order to timely detect RSV-RTI and to
  ensure cases are timely captured by the study sites, both active and passive
  surveillance will be conducted:
  - Passive surveillance: parent(s)/LAR(s) are instructed to contact the investigator/study staff as soon as the subject experiences new RTI symptoms (cough, runny nose or blocked nose) or worsening of RTI symptoms, or in case of difficulty in breathing or wheezing.
  - Active surveillance: parent(s)/LAR(s) of all the subjects will be contacted by the investigator/study staff on a regular basis (weekly during the RSV season and every month outside the RSV season) to identify any potential RSV-RTI and to remind the parent(s)/LAR(s) of the subjects to report any new occurrence of RTI symptoms (cough, runny nose or blocked nose), or in case of difficulty in breathing or wheezing as soon as possible.

Refer to Section 9.2 of the protocol for more information about active and passive surveillance.

- Surveillance for spontaneous or excessive bleeding Subjects' parent(s)/LAR(s) will be instructed to contact the investigator/study staff if their child presents symptoms of spontaneous bleeding or easy bruising or if their child develops a rash, within 30 days after either vaccination (Visit 1 and Visit 3), in order to detect any thrombocytopenic petechiae or purpura. The investigator will, based on his/her medical judgment, measure the total blood count and appropriately investigate infants with clinical suspicion of low platelets.
- **Group description**: For the <u>blinded report on safety/reactogenicity</u>, the analyses will be presented as one group (RSV groups and Placebo group being pooled).

The following group names for the unblinded analysis will be used in the TFLs, to be in line with the T-domains:

| Group<br>order in<br>tables | Group label in tables | Group definition for footnote | Pooled Groups label<br>in tables –<br>UNBLINDED<br>ANALYSIS | Pooled definition<br>for footnote -<br>UNBLINDED<br>ANALYSIS |
|---|---|---|---|---|
| 1 | RSVBEX1D | RSV 1D + BEXERO 3D | RSV 1D | Pooled 1D RSV |
| 2 | RSVNIM1D | RSV 1D +NIMENRIX 3D | | |
| 3 | RSVSYN1D | RSV 1D +SYNFLORIX 3D | | |
| 4 | RSVMEN1D | RSV 1D +MENVEO 2D | | |
| 5 | RSVPBO1D | RSV 1D + PLACEBO | | |
| 6 | RSVBEX2D | RSV 2D + BEXERO 3D | RSV 2D | Pooled 2D RSV |
| 7 | RSVNIM2D | RSV 2D +NIMENRIX 3D | | |
| 8 | RSVSYN2D | RSV 2D +SYNFLORIX 3D | | |
| 9 | RSVMEN2D | RSV 2D +MENVEO 2D | | |
| 10 | RSVPBO2D | RSV 2D + PLACEBO | | |
| 11 | BEXERO | BEXERO 3D | COMP_PLB | Pooled comparator |
| 12 | NIMENRIX | NIMENRIX 3D | | |
| 13 | SYNFLORIX | SYNFLORIX 3D | | |
| 14 | MENVEO | MENVEO 2D | | |
| 15 | PLACEBO | PLACEBO | | |

### 3. OBJECTIVES/ENDPOINTS

# 3.1. Objectives

## 3.1.1. Primary Objective

• To evaluate the safety and reactogenicity of the RSV investigational vaccine when administered IM as one (1.5x10<sup>10</sup> vp) dose or as two (5x10<sup>10</sup> vp) doses according to a 0, 1-month schedule, up to 60 days after Dose 1 (i.e., Day 61) in infants aged 6 and 7 months

## 3.1.2. Secondary Objective

- To evaluate the occurrence of RSV respiratory tract infections of any severity from Visit 1 (Day 1, after Dose 1) up to the end of the first RSV transmission season, in infants aged 6 and 7 months
- To evaluate the safety of the RSV investigational vaccine when administered IM as one (1.5x10<sup>10</sup> vp) dose or as two (5x10<sup>10</sup> vp) doses according to a 0, 1-month schedule, from study start (Day 1) up to the end of the second RSV transmission season in infants aged 6 and 7 months
- To evaluate the occurrence of RSV respiratory tract infections from Visit 1 (Day 1, after Dose 1) up to the end of the second RSV transmission season, in infants aged 6 and 7 months.

204894 (RSV-PED-011) Statistical Analysis Plan Final

- To evaluate the occurrence of very severe RSV-LRTI from Visit 1 (Day 1, after Dose 1) up to the end of the first RSV transmission season in RSV infected infants aged 6 and 7 months with a negative RSV exposure status (at screening based on instream baseline serological testing.
- To evaluate the humoral immunogenicity induced by the RSV investigational vaccine when administered IM as one (1.5x10<sup>10</sup> vp) dose or as two (5x10<sup>10</sup> vp) doses according to a 0, 1-month schedule, from study start (Day 1) up to the end of the first RSV transmission season, in infants aged 6 and 7 months.

# 3.1.3. Tertiary objective

• If deemed necessary, to further characterize the immune response of the RSV investigational vaccine when one (1.5x10<sup>10</sup> vp) dose or two (5x10<sup>10</sup> vp) doses are administered IM according to a 0, 1-month schedule to infants aged 6 and 7 months

# 3.2. Endpoints

## 3.2.1. Primary endpoints

- Occurrence of adverse events (AEs) from first vaccination (Day 1) up to Day 61
  - Occurrence of each solicited local and general AE, during a 7-day follow-up period after each vaccination (i.e., the day of vaccination and 6 subsequent days)
  - Occurrence of any unsolicited AE, during a 30-day follow-up period after each vaccination (i.e., the day of vaccination and 29 subsequent days)
  - Occurrence of any serious adverse event (SAE) from Day 1 up to Day 61
  - Occurrence of episode of spontaneous or excessive bleeding (AE of special interest), during a 30-day follow-up period after each vaccination

## 3.2.2. Secondary endpoints

- Occurrence of RSV-RTI, RSV-LRTI, severe RSV-LRTI and very severe RSV-LRTI
  (according to standardized case definitions) as from first vaccination (Day 1) up to
  the end of the first RSV transmission seasons.
- Occurrence of RSV-RTI, RSV-LRTI, severe RSV-LRTI and very severe RSV-LRTI
  (according to standardized case definitions) as from first vaccination (Day 1) up to
  the end of the second RSV transmission seasons.
- Occurrence of SAEs from first vaccination (Day 1) up to the end of the second RSV transmission seasons.
- Occurrence of RSV-LRTI (AE of special interest) as from first vaccination (Day 1)
  up to the end of the first RSV transmission season, and up to the end of the second
  RSV transmission seasons.

204894 (RSV-PED-011) Statistical Analysis Plan Final

- Occurrence of very severe RSV-LRTI (according to standardized case definitions) among RSV infected infants with a negative RSV exposure status (at screening based on in-stream baseline serological testing) from first vaccination (Day 1) up to the end of the first RSV transmission seasons.
- Humoral response to the investigational RSV vaccine, pre-vaccination (Screening), post-Dose 1 (Day 31) and post-Dose 2 (Day 61 and at the end of the first RSV transmission season):
  - Neutralizing antibody titers against RSV-A
  - RSV F antibody concentrations

### 3.2.3. Tertiary endpoints

- Humoral response to the investigational RSV vaccine, pre-vaccination (Screening), post-Dose 1 (Day 31) and post-Dose 2 (Day 61)
  - Palivizumab-competing antibody concentrations
- Any further exploratory immunology to detect disease-related or vaccine-related immune responses, such as but not limited to
  - Anti-vector immunity: neutralization

### 4. ANALYSIS SETS

### 4.1. Definition

### 4.1.1. Exposed Set

The Exposed Set (ES) will include all subjects with at least one study vaccine administration documented.

- A safety analysis based on the ES will include all vaccinated subjects.
- An immunogenicity analysis will be conducted on the ES and will include all vaccinated subjects for whom immunogenicity data are available.

The ES analysis will be performed per treatment actually administered at Dose 1

# 4.1.2. Exposed Set of subjects with a negative RSV exposure status

The Exposed Set of subjects with a negative RSV exposure status will include all vaccinated subjects assessed as RSV unexposed at screening based on in-stream baseline serological testing

The safety analysis of incidence of RSV-LRTI will be conducted on the cohort of subjects with a negative RSV exposure status (at screening based on in-stream baseline serological testing) as well as on the entire ES.

### 4.1.3. Per-protocol Set for analysis of immunogenicity

The per-protocol set (PPS) cohort for analysis of immunogenicity will be defined by timepoint (Day 31, Day 61 and End of the first RSV transmission season) and will consist of all subjects from the ES who complied with eligibility criteria, study procedures up to the end of the study and had immunogenicity results in the epoch as described below,

More specifically, the PPS cohort for analysis of immunogenicity for specific timepoint (Day 31 [Visit 3], Day 61 [Visit 5] and at end of the first RSV transmission season [Visit 7]) will include all evaluable subjects:

- Who met all eligibility criteria (i.e., no protocol violation linked to the inclusion/exclusion criteria, including age).
- Who received study vaccine as scheduled per protocol.
- For whom the administration route and site of the vaccine was as according to protocol.
- Who received the vaccine according to protocol procedures.
- Who complied with the vaccination schedule, as specified Table 4 in of the SAP.
- Who did not receive a concomitant medication/product/vaccine leading to exclusion from a PPS analysis, as described in Section 7.6.2 of the protocol, up to Day 31 (Visit 3)/up to Day 61 (Visit 5) /at Visit 7 (end of the first RSV transmission season).
- Who complied with the timings of the post vaccination blood sampling for immune response evaluation, up to Day 31 (Visit 3)/up to Day 61 (Visit 5) /at Visit 7 (end of the first RSV transmission season), as specified in Table 4 of the SAP.

When presenting different time-points, the PPS for immunogenicity will be adapted for each time-point (Day 31, Day 61 and End of first RSV transmission season).

Table 4 presents the intervals between study visits that determine subjects' eligibility for inclusion in the PPS analysis.

Table 4 Maximum allowed interval between study visits for PPS

| Interval | Allowed length of interval <sup>1</sup> |
|---|---|
| Visit 1 (Day 1) → Visit 3 (Day 31) | 23 - 44 days |
| Visit 1 (Day 1) → Visit 5 (Day 61) | 60 - 81 days |
| Visit 3 (Day 31) → Visit 5 (Day 61) | 28 - 37 days <sup>2</sup> |
| Visit 5 (Day 61) → Visit 7 | 90 days to the defined end of transmission season or |
| (end of the first RSV transmission season) | up to 4 weeks after |

<sup>&</sup>lt;sup>1</sup> Subjects will not be eligible for inclusion in the PP cohort for analysis of immunogenicity if they make the study visit outside this interval.

<sup>&</sup>lt;sup>2</sup> The interval between Visit 1 and Visit 5 must be a minimum of 60 days to be in line with the active comparator vaccination schedules as per the respective approved labels.

# 4.2. Criteria for eliminating data from Analysis Sets

Elimination codes are used to identify subjects to be eliminated from analysis. Detail is provided below for each set.

# 4.2.1. Elimination from Exposed Set (ES)

Code 1030 (Study vaccine not administered at all), code 900 (invalid informed consent) and code 800 (fraudulent data) will be used for identifying subjects eliminated from ES.

# 4.2.2. Elimination from Exposed Set (ES) subjects with a negative RSV exposure status

Code 1030 (Study vaccine not administered at all), code 900 (invalid informed consent) and code 800 (fraudulent data) will be used for identifying subjects eliminated from ES. Additionally, code 2020 (RSV- seropositive antibody status at baseline) will be used to identify all the subject with negative RSV exposure status.

# 4.2.3. Elimination from Per-protocol analysis Set (PPS)

## 4.2.3.1. Excluded subjects

A subject will be excluded from the PPS analysis under the following conditions

For codes 1040, 1070, 1080, 1090, 2040, 2060, 2070, 2080: subjects will be eliminated from a specific visit (at which the condition is met) onwards.

For codes 2090, 2100, 2120: subjects will be eliminated at the specific visit at which the condition is met

| Code | Condition under which the code is used | Visit (timepoints) where the code is applicable | Applicable for analysis set |
|---|---|---|---|
| 800 | Fraudulent data | All | All |
| 900 | Invalid informed consent | All | all |
| 1030 | Study vaccine not administered at all | All | Safety, immunology |
| 1040 | Administration of concomitant vaccine(s) forbidden in the protocol:- • Any investigational or non-registered product (drug or vaccine) other than the study vaccines used during the study period • A vaccine not foreseen by the study protocol administered during the period starting 30 days before the first dose and ending 30 days after the last dose of vaccine*, with the exception of: - Scheduled routine pediatric vaccines which may be administered ≥ 7 days before a dose and ≥ 7 days after a dose of study vaccines, with the exception of live viral vaccines which may be administered | Visit 3,5, 7 | Immunogenicity |

| Statistical Analysis | | | |
|---|---|---|---|
| Code | Condition under which the code is used | Visit (timepoints) where the code is applicable | Applicable for analysis set |
| | ≥ 14 days before a dose or ≥ 7 days after | | |
| | a dose. | | |
| | <ul> <li>Vaccines needed for urgent individual</li> </ul> | | |
| | medical need (e.g., rabies prophylaxis | | |
| 1050 | Randomisation failure | All | Immunogenicity |
| 1060 | Randomisation code was broken | All | Immunogenicity |
| 1070 | Subjects got vaccinated with the correct vaccine but | All | Immunogenicity |
| | containing a lower volume | | |
| 1070 | Vaccination not according to protocol: | All | Immunogenicity |
| | Wrong replacement or study vaccine | | |
| | administered (not compatible with the vaccine | | |
| | regimen associated to the treatment number) | | |
| | Site or route of study vaccine administration | | |
| | wrong or unknown | | |
| | <ul> <li>Administration not according to protocol for</li> </ul> | | |
| | reason specified by the investigator, other than | | |
| | side, site and route | | |
| 1080 | Vaccine temperature deviation (vaccine administered | All | Immunogenicity |
| | despite a Good Manufacturing Practices (GMP) no-go | | |
| | temperature deviation for RSV vaccines only) | | |
| 1090 | Expired vaccine administered (only applicable for RSV | All | Immunogenicity |
| 2212 | vaccine) | | |
| 2010 | Protocol violation (inclusion/exclusion criteria including | All | Immunogenicity |
| 00.10 | age) | 10000 | |
| 2040 | Administration of any medication forbidden by the | Visit 3, 5, 7 | Immunogenicity |
| | protocol: | | |
| | Any investigational or non-registered product (drug) other than the study vessions used during | | |
| | (drug) other than the study vaccines used during | | |
| | the study period | | |
| | Long-acting immune-modifying drugs<br>administered at any time during the study period | | |
| | <ul> <li>Immunosuppressants or other immune-<br/>modifying drugs administered chronically (i.e.,</li> </ul> | | |
| | more than 14 days in total) during the study | | |
| | period period | | |
| | Immunoglobulins and/or any blood products | | |
| | administered during the study period | | |
| 2050 | Underlying medical condition forbidden by the protocol | Visit 3, 5, 7 | Immunogenicity |
| 2060 | Intercurrent medical condition | Visit 3, 5, 7 | Immunogenicity |
| _000 | → Intercurrent medical condition that has the | 7,010,0,7 | |
| | capability of altering immune response, or alteration of | | |
| | initial immune status (suspected or confirmed | | |
| | immunosuppressive or immunodeficient condition) | | |
| | which may influence immune response | | |
| 2070 | Concomitant infection not related to the vaccine which | Visit 3, 5, 7 | Immunogenicity |
| | may influence immune response | , , | 0 7 |
| 2080 | Subjects did not comply with vaccination schedule:- | Visit 3 | Immunogenicity |
| | Number of days between dose 1 and dose 2 is outside | | , |
| | [23-44 days] | | |

| | Statistical Arialysis Flair | | |
|---|---|---|---|
| Code | Condition under which the code is used | Visit (timepoints) where the code is applicable | Applicable for analysis set |
| 2090 | <ul> <li>Subjects did not comply with blood sample schedule</li> <li>Number of days between dose 1 and visit 3 blood sample is outside [23-44 days]</li> <li>Number of days between dose 1 and visit 5 blood sample is outside [60-81 days]</li> <li>Number of days between dose 2 and visit 5 blood sample is outside [28-37 days] for RSV 2D group</li> <li>Number of days between visit 5 blood sample and visit 7 blood sample is outside [92-148 days]</li> </ul> | Visit 3, 5, 7 | Immunogenicity |
| 2100 | Serological results not available post-vaccination:- No immunological result at visit x for all 2 tests - RSV A Neutralising antibody titer and RSVPreF3-specific IgG antibody concentration | Visit 3, 5 and 7 | Immunogenicity |
| 2120 | Obvious incoherence or abnormality or error in data:- Incoherence between CRF and results, wrong sample labelling, Central/internal/external lab deviations; incorrect spinning/processing of sample including processing within the time required by protocol; temperature deviations from range defined in protocol and/or SPM - room temperature/refrigerator/freezer; an assessment was completed but was not completed according to protocol or SPM. | Visit 3, 5, 7 | Immunogenicity |

## 5. STATISTICAL ANALYSES

Note that standard data derivation rules and stat methods are described in "business rules document" and will not be repeated below. The study specific data derivation rules and stat methods will be described in section 9.

# 5.1. Demography

# 5.1.1. Analysis of demographics/baseline characteristics planned in the protocol

The analysis of demographics will be performed on the ES and on the PPS cohort for immunogenicity for each RSV + comparator vaccine group and each active control comparator group and also for the pooled RSV vaccine and pooled comparator group.

Demographic characteristics (age at vaccination in months, sex, country and race and vital signs), cohort description will be summarized by group using descriptive statistics:

- Frequency tables will be generated for categorical variables such as race.
- Mean, median, standard deviation and range will be provided for continuous data such as age.

The distribution of subjects will be tabulated as a whole and per group.

204894 (RSV-PED-011) Statistical Analysis Plan Final

Withdrawal status will be summarized by group using descriptive statistics:

- The number of subjects enrolled into the study as well as the number of subjects excluded from PP analyses will be tabulated.
- The numbers of withdrawn subjects will be tabulated according to the reason for withdrawal.

### 5.1.2. Additional considerations

- Summary of important protocol deviation leading to elimination will be presented. An individual listing will also be presented for this.
- Consort tables for flow of subject from enrolment to randomization and randomization to exposed will also be presented.
- The following table will be performed for web public disclosure
  - Percentage of Enrolled subjects by country will be tabulated by group,
  - Percentage of Enrolled subjects by age categories will be tabulated by group.

# 5.2. Immunogenicity

### 5.2.1. Analysis of immunogenicity planned in the protocol

The primary analysis will be performed on the PPS for immunogenicity and, if in any group the percentage of vaccinated subjects with serological results excluded from the PPS for immunogenicity is more than 10%, a second analysis will be performed on the ES. The results from immunogenicity analysis will be reported by the pooled RSV vaccine group and the pooled comparator group

For the final analysis, the Adapted PPS for immunogenicity analysis will be used which allows the summary of immunogenicity results by time point. In summary table on the Adapted PPS for immunogenicity, immunogenicity summary result at Day 31, Day 61 and end of first RSV transmission season will be presented on PPS for immunogenicity at Day 31, Day 61 and end of first RSV transmission season, respectively.

The infants are monitored for RSV infection starting from dose 1 and, therefore, immunogenicity analyses can be adjusted to exclude those infants with an infection prior to sampling.

### 5.2.1.1. Within groups assessment

## 5.2.1.1.1. Analysis of secondary objectives

For three pooled groups, at each timepoint that blood samples are collected for humoral immune response against the investigational RSV vaccine (neutralizing antibody titers against RSV-A, RSV F antibody concentrations).

- Geometric mean titers/concentrations (GMTs/GMCs) will be tabulated with 95% CI and represented graphically.
- Percentage of subjects above the sero-positivity threshold will be tabulated with exact 95% CI.
- Antibody titers/concentrations will be displayed using reverse cumulative curves.
- The distributions (< 128, 128-256, > 256-512, > 512-1024, > 1024-2048, > 2048-4096, > 4096) of neutralizing antibody titers/concentrations will be tabulated.
- Individual post-vaccination versus pre-vaccination results will be plotted using scatter plots. Results of the comparator group will be used as a reference.
- Geometric mean of ratios of antibody titers/concentrations at each post-vaccination timepoint over pre-vaccination will be tabulated with 95% CI.
- Distribution of the fold increase of the neutralizing antibody titers will be tabulated by pre-vaccination titer category.
- The kinetics of individual antibody titers/antibody concentrations results will be plotted as a function of time for subjects with results available at all timepoints.

An immunogenicity analysis will also be performed on the ES with a negative RSV exposure status (at screening based on in-stream baseline serological testing) for whom immunogenicity data are available.

At study end, an additional analysis of immunogenicity will be performed on infants by baseline values (as per the cut-off used to define RSV naïve serostatus).

### 5.2.1.1.2. Analysis of tertiary objective

If available, any further exploratory immunology results (including, but not limited to anti-vector immunity and palivizumab-competing antibody concentrations) will be reported by timepoint for the two pooled RSV vaccine groups and the pooled comparator group using descriptive summary statistics.

### 5.2.2. Additional considerations

- Summary statistics for neutralizing antibody titers against RSV-A, RSV F antibody concentrations (Minimum, Mean, median, SD, 1<sup>st</sup> quartile, 3<sup>rd</sup> quartile, Maximum) will be presented.
- Distribution of the fold increase of the neutralizing antibody titers will be tabulated by pre-vaccination titer category (percentage of subjects with a fold increase equal to

204894 (RSV-PED-011) Statistical Analysis Plan Final

or above 1, 2, 2.5, 3, 4, 6, 8 10, 11 and 12 by pre-vaccination titre category: (< 128, 128-256, > 256-512, > 512-1024, > 1024-2048, > 2048-4096, > 4096, and by cumulative category:  $<128, \ge 128, \ge 256, \ge 512, \ge 1024, \ge 2048, \ge 4096$ .). The thresholds for presentation of titres in distribution table and for fold increase will be further adjusted at Day 61 analysis as needed.

- For three pooled groups, at each timepoint that blood samples are collected for humoral immune response against the investigational RSV vaccine (neutralizing antibody titrs against RSV-A, RSV F antibody concentrations, following additional analysis will be performed on PPS by baseline values (sero-negative vs sero-positive for RSV as per cut-off defined for RSV naïve serostatus) at the end of study:-
  - Geometric mean titers/concentrations (GMTs/GMCs) will be tabulated with 95% CI and represented graphically.
  - The distributions of neutralizing antibody titers/concentrations will be tabulated.
  - Geometric mean of ratios of antibody titers/concentrations at each postvaccination timepoint over pre-vaccination will be tabulated with 95% CI
  - Summary statistics for neutralizing antibody titers against RSV-A, RSV F antibody concentrations (Minimum, Mean, median, SD, 1<sup>st</sup> quartile, 3<sup>rd</sup> quartile, Maximum) will be presented.

# 5.3. Analysis of safety and reactogenicity

# 5.3.1. Analysis of safety and reactogenicity planned in the protocol

### 5.3.1.1. Within groups assessment

The safety will be descriptively summarized based on the ES. The analysis of local AEs, general AEs and fever will be reported for each RSV + comparator vaccine group and each active control comparator group and also for the pooled RSV vaccine and pooled comparator groups. For the analysis of SAEs and AE of specific interest, the analysis will be performed only on the pooled RSV and pooled comparator groups.

The percentage of subjects with at least one local AE (solicited and unsolicited), with at least one general AE (solicited and unsolicited) and with any AE during the 7-day or 30-day follow-up period will be tabulated with exact 95% confidence interval (CI) after each vaccine dose and overall. The percentage of doses followed by at least one local AE (solicited and unsolicited), by at least one general AE (solicited and unsolicited) and by any AE during the 7-day or 30-day follow-up period will be tabulated, overall vaccination course, with exact 95% CI. The same computations will be done for Grade 3 AEs, for any AEs considered related to vaccination for any Grade 3 AEs considered related to vaccination and AEs resulting in a medically attended visit.

The percentage of subjects reporting each individual solicited local AE (any grade, Grade 2, Grade 3, resulting in a medically attended visit) and solicited general AE (any grade, Grade 2, Grade 3, any related, Grade 2 related, Grade 3 related, resulting in medically attended visit) during the 7-day follow-up period (Day 1-7) will be tabulated for each

204894 (RSV-PED-011) Statistical Analysis Plan Final

RSV + comparator vaccine group and each active control comparator group and also for the pooled RSV vaccine and pooled comparator groups after each vaccine dose and overall. Similarly, the percentage of doses followed by each individual solicited local and general AE and their sub-categories, will be tabulated, overall vaccination course, with exact 95% CI.

For fever, the number and percentage of subjects reporting fever by half degree (°C) cumulative increments during the 7-day follow-up period (Day 1-7) will be tabulated for each RSV + comparator vaccine group and each active control comparator group and also for the pooled RSV vaccine and pooled comparator groups after each vaccine dose and overall. Similar tabulations will be performed for any fever with a causal relationship to vaccination, Grade 3 (> 40.0°C) causally related fever and for any fever resulting in a medically attended visit. In addition, the prevalence of any and Grade 3 fever will be presented graphically over time after vaccination.

For clinical safety laboratory parameters, a listing of laboratory value outside the normal range for the unscheduled visits will be provided as per the toxicity scale referred in the protocol. Laboratory values will be classified according to toxicity criteria (Table 7) of the SAP.

Laboratory values that are outside the normal range will also be flagged in the data listings, along with corresponding normal ranges and assessment of clinical significance

The percentage of subjects with unsolicited AEs within 30 days (Day 1-30) after each vaccine dose (overall doses) with its exact 95% CI will be tabulated RSV + comparator vaccine group and each active control comparator group and also for the pooled RSV vaccine and pooled comparator groups and by MedDRA preferred term. Similar tabulation will be done for Grade 3 unsolicited AEs, for any causally related unsolicited AEs, for Grade 3 causally related unsolicited AEs and for unsolicited AEs resulting in a medically attended visit. The verbatim reports of unsolicited AEs will be reviewed by a physician and the signs and AEs will be coded according to the MedDRA Dictionary for Adverse Reaction Terminology. Every verbatim term will be matched with the appropriate Preferred Term.

The percentage of subject with episode of spontaneous or excessive bleeding (AE of specific interest), during a 30-day follow-up period after each vaccination will be tabulated according to associated Preferred Term code mentioned in Section 9.4 of the SAP.

The percentage of subjects with RSV-LRTI (AE of specific interest) from Dose 1 up to end of the first RSV transmission season and from Dose 1 up to end of second RSV season will be tabulated according to associated Preferred Term code presented in the Section 9.4 of the SAP.

The percentage of subjects with SAE within 30 days (Day 1-30) after each vaccine dose with its exact 95% CI will be tabulated and by MedDRA preferred term. Similar tables will be generated for SAEs from Dose 1 to end of first RSV season and from Dose 1 to end of the second RSV season.

204894 (RSV-PED-011) Statistical Analysis Plan Final

SAEs reported throughout the study and AE of special interest will be described in detail.

The percentage of subjects using concomitant medication (any medication, any antipyretic and any antipyretic taken prophylactically, respectively) during the 7-day follow-up period (Day 1-7) and during the 30-day follow-up period (Day 1-30) will be summarized by the pooled RSV vaccine and pooled comparator groups after each vaccine dose and overall

### 5.3.1.2. Between groups assessment

Exploratory comparisons between the pooled RSV vaccine group and the pooled comparator group will be done in terms of the percentage of subjects, overall doses, reporting any Grade 2/3 AE during the 7-day follow-up period (Day 1-7) after vaccination, and/ or any fever >39.0°C during the 7-day follow-up period (Day 1-7) after vaccination, and/ or any vaccine-related SAE during the 7-day follow-up period (Day 1-7) after vaccination.

The standardized asymptotic 95% CI for the difference between the pooled RSV group and (minus) the pooled comparator group will be computed.

The standardized asymptotic 95% CI for the following differences will be computed:

- RSV1D minus COMP PLB
- RSV2D minus COMP PLB

### 5.3.2. Additional considerations

Descriptive summary of the number of days with solicited local/general adverse event during the 7 day (Days 1-7) post-vaccination period will be presented.

Percentage of subjects reporting fever (any and grade 3) and other solicited general adverse events (any grade, grade 2,3 and grade 3) during the 7-day (Days 1-7) post-vaccination period by maximum intensity will be presented in figure.

Percentage of subjects reporting solicited local adverse events (any grade, grade 2,3 and grade 3) during the 7-day (Days 1-7) post-vaccination period by maximum intensity will be presented in figure.

## 5.3.2.1. Combined Solicited and Unsolicited Adverse Events

A summary of subjects with all combined solicited (regardless of their duration) and unsolicited adverse events will be provided. Solicited adverse events will be coded by MedDRA as per the following codes

| Solicited symptom | Lower level term name | Lower level term code | Corresponding Primary Term code |
|---|---|---|---|
| Pain | Pain | 10033371 | 10033371 |
| Redness | Erythema | 10015150 | 10015150 |
| Swelling | Swelling | 10042674 | 10042674 |
| Drowsiness | Drowsiness | 10013649 | 10013649 |
| Fever | Fever | 10016558 | 10016558 |
| Irritability/Fussiness | Irritability | 10022998 | 10022998 |
| Loss of appetite | Appetite lost | 10003028 | 10003028 |

For clintrial.gov and EudraCT posting purposes, a summary of combined solicited and unsolicited non-serious adverse events will be produced by System Organ Class and preferred terms and according to occurrence of each event.

### 5.3.2.2. Exclusion of implausible solicited Adverse Event

Some local and systemic adverse events will be directly measured by the subject and will not be subject to a reconciliation process, even if they are biologically implausible. Therefore, these implausible measurements will be removed from the analysis but included in listings. Implausible measurements are summarized in the table below:

Table 5 Implausible Solicited Adverse Events

| Parameter | Implausible measurements |
|------------------|----------------------------------|
| Body temperature | ≤ 33°C or ≥ 42°C |
| Swelling | For subjects < 6 years: ≥ 250 mm |
| | Measurements < 0 mm |

### 5.3.2.3. Solicited Adverse Events

All analyses will be based on the 'as treated' analysis set. Solicited adverse events will be reported daily during the 7-day (from Day 1 to Day 7) follow up period after each vaccination, using structured diaries.

In order to summarize the data, the maximum intensity of local injection site redness/swelling (in mm) and fever (in °C) will be categorized as follows:

| Grading | Redness/swelling | Fever |
|---------|------------------|-----------------------------------------|
| 0: | None | < 38.0°C (100.4°F) |
| 1: | <5 mm | ≥ 38.0°C (100.4°F) - ≤ 39.0°C (102.2°F) |
| 2: | > 5 - ≤ 20 mm | > 39.0°C (102.2°F) - ≤ 40.0°C (104.0°F) |
| 3: | > 20 mm | > 40.0°C (104.0°F) |

204894 (RSV-PED-011) Statistical Analysis Plan Final

Fever is defined as temperature  $\geq 38.0^{\circ}\text{C} / 100.4^{\circ}\text{F}$  (regardless of the location of measurement). The preferred location for measuring temperature in this study will be the oral cavity. Body temperature will also be summarized by 0.5°C increments as follows:  $\geq 38.0, \geq 38.5, \geq 39.0, \geq 39.5, \geq 40.0$ °C.

For each of the time points or time intervals presented in the summaries, only subjects with at least one plausible observation (i.e., any non-missing values but excluding "Not done/unknown" and implausible values) for the solicited adverse events in the interval of interest will be considered. Subjects without plausible data (i.e. missing values or reported as "Not done/unknown" and implausible values) will be removed from the denominator to prevent a downward bias (towards zero).

### 5.3.2.4. Unsolicited Adverse Events

All the unsolicited adverse events occurring during the study, judged either as related, or not related to vaccination by the investigator, will be recorded. All the unsolicited adverse events/AE of specific interest (Spontaneous or excessive bleeding) occurring during the 30-day (Day 1 to Day 30) follow up period after each vaccination, and all serious adverse events/AE of specific interest (RSV LRTI) occurring from Dose 1 up to study end will be recorded according to the protocol-specified reporting rules. The original verbatim terms used by investigators to identify adverse events in the CRFs will be mapped to preferred terms using the MedDRA dictionary. The unsolicited adverse events will then be grouped by MedDRA preferred terms into frequency tables according to system organ class. Adverse events judged by the investigator as at least possibly related to study vaccine will be summarized by vaccine group, according to system organ class and preferred term within system organ class. When an unsolicited adverse event occurs more than once for a subject, the maximal severity and strongest relationship to the vaccine group will be counted.

Only vaccine-emergent adverse events will be analyzed, i.e., excluding those after a subject has given informed consent but before vaccination. The selection of unsolicited adverse events and the assignment to time intervals will be done by day of onset and not by days ongoing/persisting.

The analysis of unsolicited adverse events during the 30-day post vaccination period includes the following categories:

- Any unsolicited adverse event.
- Possibly related unsolicited adverse events.
- Grade 3 unsolicited adverse events
- Grade 3 related unsolicited adverse events.
- Serious adverse events (SAEs)
- Possibly related SAEs.
- Medically attended adverse events
- AE of specific interest (spontaneous or excessive bleeding)

SAE and AE of specific interest (RSV-LRTI) has to be reported from Day 1 up to Day 61, from Day 1 to end of 1<sup>st</sup> RSV season and from Day 1 to end of 2<sup>nd</sup> RSV season.

# 5.4. Analysis of RTI and LRTI

## 5.4.1. Analysis of RTI and LRTI planned in protocol

The primary analysis will be performed on the ES of subjects with a negative RSV exposure status (at screening based on in-stream baseline serological testing) in the pooled single dose RSV vaccine group, the pooled two dose RSV vaccine group, and the pooled comparator group separately for first and second RSV seasons and overall. A similar analysis will be performed on the entire ES. As primary analysis, the assessment of RSV infection will be performed using the quantitative RT-PCR according to standardized case definitions (see Table 6 of the SAP) based on the available WHO case definitions.

The number of RSV infections within each group and the maximum disease severity of the event will be tabulated. The rate (with 95% CI) of RSV-RTI and RSV-LRTI and infections progressing to hospitalization will be evaluated for each of the three pooled groups.

The rate of very severe RSV-LRTI among RSV infected infants with a negative RSV exposure status (at screening based on in-stream baseline serological testing) from first vaccination (Day 1) up to the end of the first RSV transmission season will be estimated as well as 95% one-sided lower CI.

The proportion and the relative risk of subjects with at least one RSV-associated RTI (with 95% CI) between each of two pooled RSV vaccine groups and the pooled control group will be calculated for both the cohort of subjects with a negative RSV exposure status (at screening based on in-stream baseline serological testing) on the ES and on the entire ES. The same descriptive analysis will be performed for subjects with at least one RSV-associated LRTI and those with at least one RSV-associated severe LRTI.

Descriptive analyses (mean, median, min, max) of viral load assessed by the quantitative RT-PCR (RSV-A/B) of all cases as listed in Table 6 of the SAP will be tabulated by case category. This analysis will also be done on the three pooled groups.

The incidence rate of all cases as listed in Table 6 of the SAP (with 95% CI) will be calculated by the three pooled groups. The same descriptive analysis will be performed for all cause LRTI and all cause severe LRTI. These will also be presented for each viral etiology identified by the multiplex PCR.

The incidence rate of asymptomatic RSV infections (with 95% CI) detected by the quantitative PCR (RSV-A/B), will be tabulated by the three pooled groups. Descriptive analyses (mean, median, min, max) of viral load assessed by the quantitative RT-PCR (RSV-A/B) of those asymptomatic RSV infections will also be done on the three pooled groups.

The RVP (Multiplex PCR) on specimens from all RSV-A/B positive and confirmed LRTI cases, according to case definition presented in Table 6 (Figure 3 of the protocol for the decision tree), will be tabulated as a qualitative assessment profiling the potential coinfections occurring in these subjects.

### 5.4.2. Additional consideration

In addition to above planned analysis for RTI and LRTI, following additional analysis is planned: -

- Descriptive analysis on maximum viral load per subject based on qRT-PCR confirmed RSV infection of maximum severity will be performed.
- Listing will be presented for all cases of RSV infection at Day 731 with the details of gender, age at episode, country, site, day of event (i.e days since first visit), classification according to maximum severity of episode as RSV RTI/RSV LRTI/RSV severe LRTI and RSV very severe LRTI, RSV hospitalization 'Yes/No', SpO2 value, respiratory rate, result of RSV qRT-PCR and RVP result will be presented.
- Listings will be generated at Day 731 for all hospitalized cases with gender, age at
  episode, classification according to maximum severity of episode as (RSV RTI/RSV
  LRTI/ RSV severe LRTI and RSV very severe LRTI), RVP result, total number of
  calendar days on which the child was hospitalized, days requiring
  monitoring/nursing observation, days requiring nasogastric or intravenous fluids,
  days requiring supplemental oxygen, days requiring respiratory support excluding
  mechanical ventilation, days requiring mechanical ventilation and days requiring
  pediatric intensive care unit management.

## 6. ANALYSIS INTERPRETATION

For the occurrence of very severe RSV-LRTI among RSV infected infants with a negative RSV exposure status (at screening based on in-stream baseline serological testing) from first vaccination (Day 1) up to the end of the first RSV transmission season, if the upper boundary of the 95% one-sided lower CI of the rate is under 80%, it indicates that the very severe RSV-LRTI rate is less than that of the historic RSV-FI trials [Kim, 1969].

Comparative analyses will be exploratory and should be interpreted with caution considering that there is no adjustment for multiplicity and that group sizes are small for these comparisons.

### 7. CONDUCT OF ANALYSES

# 7.1. Sequence of analyses

The statistical analyses will be performed in 3 steps:

• An analysis will be performed when all data up to Day 61 are available. Additional safety data available at the time of this analysis will be described. At this point, the statistician will be unblinded (i.e., individual subject treatment assignments will be available) and the study will be conducted in a single blind manner, with patients remaining blinded up to the last study visit (end of the second RSV transmission season). Summary results may unblind some specific subjects, but no individual listings will be provided and the investigator will not have access to the treatment
204894 (RSV-PED-011) Statistical Analysis Plan Final

allocation up to the last study visit (end of the second RSV transmission season), except in case of emergency unblinding (see Section 9.8 of the protocol)

- An analysis will be performed when all data up to Visit 7 (end of the first RSV transmission season, i.e., data that are as clean as possible) are available. No individual listings will be provided.
- The final analysis will be performed when all data up to study conclusion (end of the second RSV transmission season) are available. An integrated clinical study report containing all data will be written and made available to the investigators at that time.

If the data for tertiary endpoints become available at a later stage, (an) additional analysis/ analyses will be performed. These data will be documented in annex(es) to the study report and will be made available to the investigators at that time.

| Description | Disclosure Purpose<br>(CTRS=public posting, SR=study report, internal) |
|---|---|
| Day 61 analysis | Internal, web disclosure |
| End of RSV season 1 | Internal |
| End of RSV season 2 | Web disclosure, Study report |

# 7.2. Statistical considerations for interim analyses

No interim analyses are planned

## 8. CHANGES FROM PLANNED ANALYSES

Following are few changes from planned analysis:-

- In the protocol, we have PPS up to Day 61 which included Day 31 as well. To have better clarity with respect to PPS for Day 31, the text has been re-worded for the definition of PPS population. PPS has also been defined for Day 31 timepoint along with PPS at Day 61 and end of 1<sup>st</sup> RSV transmission season. Also, as the timepoint 'End of 1<sup>st</sup> RSV transmission season is not exactly Day 365, so the Day 365 has been removed and only kept as PPS at end of 1<sup>st</sup> RSV transmission season. The criteria of eliminating subject from the PPS of respective timepoint is accordingly reworded.
- In the protocol amendment 3, it is mentioned under Analysis of Immunogenicity section that 'In summary table on the Adapted PPS for immunogenicity, PPS for immunogenicity at Day 61 will be used for Pre, Day 31 and Day 61 immunogenicity summary and PPS for immunogenicity at Day 365 for Day 365 immunogenicity summary.' As we have added the PPS for Day 31 in the SAP, accordingly the summary table presentation has been modified as 'In summary table on the Adapted PPS for immunogenicity, immunogenicity summary result at Day 31, Day 61 and end of first RSV transmission season) will be based on PPS of Day 31, Day 61 and end of first RSV transmission season, respectively'.
- Table to present percentage of responders in terms of neutralizing antibody titers with 95% CI has been removed as there is no definition of response available.

# 9. NON-STANDARD DATA DERIVATION RULES AND STATISTICAL METHODS

The following sections describe additional derivation rules and statistical methods which are not presented in section 10.1 (Business rules for standard data derivations and statistical methods).

# 9.1. Immunogenicity

• Assay cut-off for the humoral immunity will be per the following table

| Component | Method | Unit | Cut-off |
|---|---|---|---|
| Respiratory Syncytial Virus A Ab | NEUTRALIZATION | ED60 | 18 |
| Respiratory Syncytial Virus F protein Ab.lgG (Anti-RSV PreF antibody) | ELISA | EU/ml | 10 |
| Respiratory Syncytial Virus F protein Ab.lgG (Palivizumab competing Ab) | ELISA | μg/ml | 9.6 |

- For RSV neutralizing assay, the LLOQ and ULOQ is set at 18ED60 and 21654 ED60. For analysis, the cut-off is set at the lower limit of quantification. For results below the cut-off, an arbitrary value of half of the cut-off will be considered for calculation of GMC and fold increase. The result above the ULOQ is set at ULOQ for analysis.
- For anti-RSV PreF antibody and RSV PCA, the cut-off is set at the level of detection. For results below the cut-off (LOD), an arbitrary value of half of the cutoff will be considered for calculation of GMC and fold increase.

#### 9.2. RTI and LRTI

During the analysis of the study, all cases identified during the surveillance of RSV-RTI will be definitively classified as either RTI, LRTI, severe LRTI or very severe LRTI according to the standardized case definitions (Table 6 in the SAP) based on the available World Health Organization (WHO) case definitions (Table 6 in the protocol)

Table 6 Case definitions for data analysis

| Case | At sea level up to 2500 meters elevation | Above 2500 meters elevation |
|---|---|---|
| RSV-RTI | Runny nose OR blocked nose OR cough | Same |
| | AND | |
| | Confirmed RSV infection <sup>4</sup> | |
| RSV-LRTI | History of cough OR difficulty breathing <sup>1</sup> | Same but with |
| | AND | SpO2 <92% |
| | SpO <sub>2</sub> < 95% <sup>2</sup> , OR RR increase <sup>3</sup> | |
| | AND | |
| | Confirmed RSV infection <sup>4</sup> | |
| severe RSV- | Meeting the case definition of RSV-LRTI | Same but with |
| LRTI | AND | SpO2 <90% |
| | SpO <sub>2</sub> < 93% <sup>2</sup> , OR lower chest wall in-drawing | ' |
| very severe | Meeting the case definition of RSV-LRTI | Same but with |
| RSV-LRTI | AND | SpO2 <88% |
| | SpO <sub>2</sub> < 90% <sup>2</sup> , OR inability to feed, OR failure to respond / unconscious | - |

| Case | At sea level up to 2500 meters elevation | Above 2500 meters elevation |
|---|---|---|
| RSV | Confirmed RSV infection 5 | Same |
| hospitalization | AND | |
| _ | Hospitalized for acute medical condition <sup>6</sup> | |
| All-cause LRTI | History of cough OR difficulty breathing 1 | Same but with |
| | AND | SpO2 <92% |
| | SpO <sub>2</sub> < 95% <sup>2</sup> , OR RR increase <sup>3</sup> | - |

**LRTI** = lower respiratory tract infections; **RR** = respiratory rate; **RTI** = respiratory tract infections; **SpO2** = blood oxygen saturation.

- For the analysis of RTI episode, a new RTI episode will be defined as any occurrence of cough, runny nose, blocked nose, wheezing or difficulty breathing with an interval of at least 7 symptom free days since the last episode of RTI that was diagnosed.
- For molecular biology (qRT-PCR test), the following cut-off will be applied: -

| System | Component | Method | Unit | Cut-off |
|---|---|---|---|---|
| Nasal swab | RSV-A RNA | Quantitative real-time PCR (qRT-PCR) | Copies/ml | 1.12 X 10 <sup>3</sup> |
| Nasal swab | RSV-B RNA | Quantitative real-time PCR (qRT-PCR) | Copies/ml | 1.47 x 10 <sup>3</sup> |

# 9.3. Hematology and Biochemistry parameters

The grading of the hematology and biochemistry lab result will be done as per the toxicity grading scales provided in the Table 7 below (Table 28 of the protocol).

Table 7 Toxicity grading scales for hematology and biochemistry parameters applicable for this study

| Component | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Hemoglobin (g/dL) | 9.0 to < 10.5 | 8.0 to < 9.0 | 7.0 to < 8.0 | < 7.0 |
| Leukocytes (cell/mm³) | 2500 to < 3500 | 1500 to < 2500 | 1000 to < 1500 | < 1000 |
| Absolute neutrophil count (cell/mm³) | 1000 to < 1300 | 750 to < 1000 | 500 to < 750 | < 500 |
| Absolute lymphocyte count (cell/mm³) | 600 to < 650 | 500 to < 600 | 350 to < 500 | < 350 |
| Platelets (cell//mm <sup>3</sup> ) | 75000 to < 150000 | 50000 to < 75000 | 25000 to < 50000 | < 25000 |
| Alanine Aminotransferase (increase by factor) | 1.1 to < 2.0 xULN | 2.0 to < 3.0 xULN | 3.00 to ≤ 8.0 xULN | > 8.0 xULN |
| Aspartate Aminotransferase (increase by factor) | 1.1 to < 2.0 xULN | 2.0 to < 3.0 xULN | 3.00 to ≤ 8.0 xULN | > 8.0 xULN |
| Creatinine (mg/dL) | 0.6 to < 0.9 | 0.9 to < 1.2 | 1.2 to ≤ 1.5 | > 1.5 |

ULN: upper limit of normal.

<sup>&</sup>lt;sup>1</sup> Based on history reported by parents.

<sup>&</sup>lt;sup>2</sup> The lowest value during the course of illness will be used.

 $<sup>^3</sup>$  RR increase defined as: $\geq$  50/minute (2 to 11 months of age);  $\geq$  40/minute (12 months of age or above); The highest value during the course of the illness will be used.

<sup>&</sup>lt;sup>4</sup> RSV infection confirmed on nasal swab positive for RSV A or B by quantitative Reverse Transcription Polymerase Chain Reaction (gRT-PCR).

<sup>&</sup>lt;sup>5</sup> RSV sampling and testing is based on medical judgment of medical practitioner or driven by algorithm.

<sup>6</sup> Hospitalization is defined as a medical decision that the infant requires admission for observation or treatment.

# 9.4. Coding for the AE of specific interest

Any of the below listed preferred term reported as an Expedited Adverse Event must be immediately escalated to the CRDL or Central Safety Physician to assess or confirm the need for an urgent IDMC review.

The list of preferred terms and associated PT codes is given below:

# **HAEMATOMA**

| Preferred term | PT code |
|------------------------------------|----------|
| abdominal wall haematoma | 10067383 |
| administration site haematoma | 10075100 |
| adrenal haematoma | 10059194 |
| aortic intramural haematoma | 10067975 |
| application site haematoma | 10068317 |
| arterial intramural haematoma | 10074971 |
| auricular haematoma | 10003797 |
| basal ganglia haematoma | 10077031 |
| brain stem haematoma | 10073230 |
| breast haematoma | 10064753 |
| broad ligament haematoma | 10006375 |
| bursal haematoma | 10077818 |
| catheter site haematoma | 10055662 |
| cephalhaematoma | 10008014 |
| cerebellar haematoma | 10061038 |
| cerebral haematoma | 10053942 |
| cervix haematoma uterine | 10050020 |
| chest wall haematoma | 10076597 |
| colonic haematoma | 10009996 |
| deep dissecting haematoma | 10074718 |
| extradural haematoma | 10015769 |
| eyelid haematoma | 10064976 |
| haematoma | 10018852 |
| haematoma evacuation | 10060733 |
| haematoma infection | 10051564 |
| hepatic haematoma | 10019676 |
| incision site haematoma | 10059241 |
| infusion site haematoma | 10065463 |
| injection site haematoma | 10022066 |
| instillation site haematoma | 10073609 |
| intestinal haematoma | 10069829 |
| intra-abdominal haematoma | 10056457 |
| intracerebral haematoma evacuation | 10062025 |

| Preferred term | PT code |
|----------------------------------|----------|
| intracranial haematoma | 10059491 |
| intraocular haematoma | 10071934 |
| laryngeal haematoma | 10070885 |
| lip haematoma | 10066304 |
| mediastinal haematoma | 10049941 |
| medical device site haematoma | 10075577 |
| mesenteric haematoma | 10071557 |
| nasal septum haematoma | 10075027 |
| oesophageal intramural haematoma | 10077486 |
| oral mucosa haematoma | 10074779 |
| ovarian haematoma | 10033263 |
| paranasal sinus haematoma | 10069702 |
| pelvic haematoma | 10054974 |
| penile haematoma | 10070656 |
| perineal haematoma | 10034520 |
| periorbital haematoma | 10034544 |
| periosteal haematoma | 10077341 |
| perirenal haematoma | 10049450 |
| peritoneal haematoma | 10058095 |
| pharyngeal haematoma | 10068121 |
| post procedural haematoma | 10063188 |
| pulmonary haematoma | 10054991 |
| renal haematoma | 10038459 |
| retroperitoneal haematoma | 10058360 |
| scrotal haematoma | 10039749 |
| spinal cord haematoma | 10076051 |
| spinal epidural haematoma | 10050162 |
| spinal subdural haematoma | 10050164 |
| splenic haematoma | 10041646 |
| spontaneous haematoma | 10065304 |
| subarachnoid haematoma | 10076701 |
| subcutaneous haematoma | 10042345 |
| subdural haematoma | 10042361 |
| subgaleal haematoma | 10069510 |
| subretinal haematoma | 10071935 |
| tongue haematoma | 10043959 |
| uterine haematoma | 10063875 |
| vaccination site haematoma | 10069472 |
| vaginal haematoma | 10046909 |
| vitreous haematoma | 10071936 |
| vulval haematoma | 10047756 |

# **HAEMORRHAGE**

| Preferred term | PT code |
|----------------------------------------|----------|
| abdominal wall haemorrhage | 10067788 |
| acute haemorrhagic conjunctivitis | 10067817 |
| administration site haemorrhage | 10075101 |
| adrenal haemorrhage | 10001361 |
| anal haemorrhage | 10049555 |
| anastomotic haemorrhage | 10056346 |
| angina bullosa haemorrhagica | 10064223 |
| application site haemorrhage | 10072694 |
| arterial haemorrhage | 10060964 |
| basal ganglia haemorrhage | 10067057 |
| bone marrow haemorrhage | 10073581 |
| brain stem haemorrhage | 10006145 |
| brain stem microhaemorrhage | 10071205 |
| breast haemorrhage | 10006254 |
| bronchial haemorrhage | 10065739 |
| catheter site haemorrhage | 10051099 |
| central nervous system haemorrhage | 10072043 |
| cerebellar haemorrhage | 10008030 |
| cerebellar microhaemorrhage | 10071206 |
| cerebral haemorrhage | 10008111 |
| cerebral microhaemorrhage | 10067277 |
| cervix haemorrhage uterine | 10050022 |
| ciliary body haemorrhage | 10057417 |
| conjunctival haemorrhage | 10010719 |
| diverticulitis intestinal haemorrhagic | 10013541 |
| diverticulum intestinal haemorrhagic | 10013560 |
| duodenitis haemorrhagic | 10013865 |
| ear haemorrhage | 10014009 |
| encephalitis haemorrhagic | 10014589 |
| gastric haemorrhage | 10017788 |
| gastroduodenal haemorrhage | 10053768 |
| gastrointestinal haemorrhage | 10017955 |
| genital haemorrhage | 10061178 |
| haemarthrosis | 10018829 |
| haematemesis | 10018830 |
| haematochezia | 10018836 |
| haematotympanum | 10063013 |
| Haematuria | 10018867 |
| haemorrhage | 10055798 |
| haemorrhage coronary artery | 10055803 |

| Preferred term | PT code |
|------------------------------------|----------|
| haemorrhage intracranial | 10018985 |
| haemorrhage subcutaneous | 10018999 |
| haemorrhage subepidermal | 10019001 |
| haemorrhage urinary tract | 10055847 |
| haemorrhagic anaemia | 10052293 |
| haemorrhagic diathesis | 10062713 |
| haemorrhagic disorder | 10019009 |
| haemorrhagic infarction | 10019013 |
| haemorrhagic ovarian cyst | 10060781 |
| haemorrhagic pneumonia | 10077933 |
| haemorrhagic thyroid cyst | 10072256 |
| haemorrhagic urticaria | 10059499 |
| injection site haemorrhage | 10022067 |
| internal haemorrhage | 10075192 |
| intestinal haemorrhage | 10059175 |
| intra-abdominal haemorrhage | 10061249 |
| intraventricular haemorrhage | 10022840 |
| iris haemorrhage | 10057418 |
| joint microhaemorrhage | 10077666 |
| lacrimal haemorrhage | 10069930 |
| large intestinal haemorrhage | 10052534 |
| laryngeal haemorrhage | 10065740 |
| lip haemorrhage | 10049297 |
| lower gastrointestinal haemorrhage | 10050953 |
| lymph node haemorrhage | 10074270 |
| mediastinal haemorrhage | 10056343 |
| mesenteric haemorrhage | 10060717 |
| mouth haemorrhage | 10028024 |
| mucocutaneous haemorrhage | 10076048 |
| mucosal haemorrhage | 10061298 |
| muscle haemorrhage | 10028309 |
| myocardial haemorrhage | 10048849 |
| naevus haemorrhage | 10062955 |
| ocular retrobulbar haemorrhage | 10057571 |
| oesophageal haemorrhage | 10030172 |
| optic disc haemorrhage | 10030919 |
| optic nerve sheath haemorrhage | 10030941 |
| ovarian haemorrhage | 10065741 |
| pancreatic haemorrhage | 10033625 |
| papillary muscle haemorrhage | 10059164 |
| parathyroid haemorrhage | 10059051 |

| Preferred term | PT code |
|------------------------------------|----------|
| parotid gland haemorrhage | 10051166 |
| pelvic haemorrhage | 10063678 |
| penile haemorrhage | 10034305 |
| pericardial haemorrhage | 10034476 |
| periorbital haemorrhage | 10071697 |
| peritoneal haemorrhage | 10034666 |
| Petechiae | 10034754 |
| pharyngeal haemorrhage | 10034827 |
| pituitary haemorrhage | 10049760 |
| post procedural haemorrhage | 10051077 |
| procedural haemorrhage | 10071229 |
| prostatic haemorrhage | 10036960 |
| pulmonary alveolar haemorrhage | 10037313 |
| pulmonary haemorrhage | 10037394 |
| putamen haemorrhage | 10058940 |
| rectal haemorrhage | 10038063 |
| renal haemorrhage | 10038460 |
| respiratory tract haemorrhage | 10038727 |
| retinal haemorrhage | 10038867 |
| retroperitoneal haemorrhage | 10038980 |
| scleral haemorrhage | 10050508 |
| skin haemorrhage | 10064265 |
| small intestinal haemorrhage | 10052535 |
| soft tissue haemorrhage | 10051297 |
| spermatic cord haemorrhage | 10065742 |
| spinal cord haemorrhage | 10048992 |
| spinal epidural haemorrhage | 10049236 |
| spinal subarachnoid haemorrhage | 10073564 |
| spinal subdural haemorrhage | 10073563 |
| splenic haemorrhage | 10041647 |
| spontaneous haemorrhage | 10074557 |
| subarachnoid haemorrhage | 10042316 |
| subdural haemorrhage | 10042364 |
| testicular haemorrhage | 10051877 |
| thalamus haemorrhage | 10058939 |
| thoracic haemorrhage | 10062744 |
| thyroid haemorrhage | 10064224 |
| tongue haemorrhage | 10049870 |
| tracheal haemorrhage | 10062543 |
| upper gastrointestinal haemorrhage | 10046274 |
| ureteric haemorrhage | 10065743 |

| Preferred term | PT code |
|------------------------------|----------|
| urethral haemorrhage | 10049710 |
| urinary bladder haemorrhage | 10046528 |
| urogenital haemorrhage | 10050058 |
| uterine haemorrhage | 10046788 |
| vaccination site haemorrhage | 10069475 |
| vaginal haemorrhage | 10046910 |
| venous haemorrhage | 10065441 |
| vitreous haemorrhage | 10047655 |
| vulval haemorrhage | 10063816 |

# **THROMBOCYTOPENIA**

| Preferred term | PT code |
|---------------------------|----------|
| bleeding time abnormal | 10049227 |
| bleeding time prolonged | 10005140 |
| coagulation test abnormal | 10063557 |
| platelet count abnormal | 10035526 |
| platelet count decreased | 10035528 |
| platelet disorder | 10035532 |
| platelet dysfunction | 10073391 |
| Thrombocytopenia | 10043554 |
| thrombocytopenic purpura | 10043561 |

# LOWER RESPIRATORY TRACT INFECTION

| Preferred term | PT code |
|-------------------------------------------|----------|
| atypical pneumonia | 10003757 |
| Bronchitis | 10006451 |
| bronchitis viral | 10053160 |
| haemorrhagic pneumonia | 10077933 |
| lower respiratory tract infection | 10024968 |
| lower respiratory tract infection viral | 10065188 |
| lung infection | 10061229 |
| Pneumonia | 10035664 |
| pneumonia respiratory syncytial viral | 10035732 |
| pulmonary sepsis | 10051739 |
| respiratory syncytial virus bronchiolitis | 10038718 |
| respiratory syncytial virus bronchitis | 10069811 |
| respiratory tract infection | 10062352 |
| respiratory tract infection viral | 10062106 |

#### 10. ANNEXES

As the SAP and TFL TOC has been developed using the old template and process, we will not have TFL as annex to this SAP. All the template applicable to the study has been added in the SAP in Section 13.

# 10.1. Business rules for standard data derivations and statistical methods

# 10.1.1. Attributing events to vaccine doses

The dose relative to an event is the most recent study dose given to a subject prior to the start of a given event. For example, if the start date of an adverse event is between Dose 1 and Dose 2, the relative dose will be Dose 1.

If an event starts on the same day as a study dose, the relative dose will be derived from the additional information provided in the CRF using the contents of the flag indicating if the event occurred before or after vaccination. If 'after vaccination' is selected, the relative dose for the event will be the one administered on the start day of the event. If 'before vaccination' is selected, the relative dose for the event will be the dose prior to this one

## 10.1.2. Handling of missing data

#### 10.1.2.1. Dates

When partially completed dates (i.e. with missing day or month) are used in calculations, the following standard rules will be applied:

- A missing day will be replaced by 15
- A missing day and month will be replaced by June 30<sup>th</sup>.

The following exceptions apply:

- Adverse event start dates with missing day:
  - If the event starts in the same month as at least one of the study doses, the contents of AE.AESTRTPT (the flag indicating if the event occurred before or after vaccination) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the first (or only) study dose given during that month. If 'before vaccination' is selected, the imputed date will be one day before the first (or only) study dose given during that month.
- Adverse event start dates with missing day and month:
  - If the event starts in the same year as at least one of the study doses, the contents of AE.AESTRTPT (the flag indicating if the event occurred before or after vaccination) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the first (or only) study dose given during that

204894 (RSV-PED-011) Statistical Analysis Plan Final

year. If 'before vaccination' is selected, the imputed date will be one day before the first (or only) study dose given during that year.

All other cases of incomplete AE or concomitant medication/vaccination start date will follow the standard rules above.

# 10.1.2.2. Laboratory data

Missing laboratory results (including immunological data) will not be replaced.

# 10.1.2.3. Daily recording of solicited symptoms

## 10.1.2.3.1. Studies with paper diaries

For studies using paper diaries which have questions in the CRF indicating the presence or absence of solicited symptoms, the following rules are applicable.

Denominators for the summary of local (or general) solicited symptoms will be calculated using the number of subjects who respond "Yes" or "No" to the question concerning the occurrence of local (or general) symptoms.

When a specific symptom is marked as having not occurred following a specific vaccination (i.e. SDTM CE.CEOCCUR=N for the specified post-vaccination period for the symptom in question), all daily measurements will be imputed as Grade 0.

When a specific symptom is marked as having occurred following a specific vaccination (i.e. SDTM CE.CEOCCUR=Y for the specified post-vaccination period for the symptom in question), any missing daily recordings will be given imputed values to allow them to contribute to the 'Any' rows but not to specific grade rows of the symptom summary tables.

When the occurrence of a specific symptom is not present (i.e. SDTM CE.CEOCCUR is neither Y nor N for the specified post-vaccination period for the symptom in question) but the group of symptoms (local or general) is marked as having occurred (i.e. SDTM CE.CEOCCUR=Y), all missing daily recordings will be given imputed values to allow them to contribute to the 'Any' rows but not to specific grade rows of the symptom summary tables.

The following table shows how subjects contribute to each category for a specific solicited symptom over the Day X to Day Y post-vaccination period:

| Solicited symptom category | Subjects included in the calculation of the numerator |
|---|---|
| Any | All subjects with at least one occurrence of the symptom at grade 1, grade 2, or grade 3 between Day X and Day Y or with the symptom marked as present and at least one missing daily recording between Day X and Day Y |
| At least grade 1 | All subjects with at least one occurrence of the symptom at grade 1, grade 2, or grade 3 between Day X and Day Y |
| At least grade 2 | All subjects with at least one occurrence of the symptom at grade 2 or grade 3 between Day X and Day Y |
| At least grade 3 | All subjects with at least one occurrence of the symptom at grade 3 between Day X and Day Y |

#### 10.1.2.4. Unsolicited adverse events

Missing severity, relationship with study vaccine, and outcome of unsolicited adverse events will not be replaced and will appear as 'UNKNOWN' in all statistical output.

#### 10.1.3. Data derivation

#### 10.1.3.1. Age at vaccination in days

When age at vaccination is to be displayed in days, it will be calculated as:

Age = date of vaccination minus date of birth

#### 10.1.3.2. Age at vaccination in months

When age at vaccination is to be displayed in months, it will be calculated as the number of complete calendar months between the date of birth (DOB) and the date of vaccination. For example:

DOB = 10JUN2017, Date of vaccination = 09JUL2018 -> Age = 12 months DOB = 10JUN2017, Date of vaccination = 10JUL2018 -> Age = 13 months

## 10.1.3.3. Age at vaccination in years

When age at vaccination is to be displayed in years, it will be calculated as the number of complete calendar years between the date of birth and the date of vaccination. For example:

DOB = 10SEP1983, Date of vaccination = 09SEP2018 -> Age = 34 years DOB = 10SEP1983, Date of vaccination = 10SEP2018 -> Age = 35 years

## 10.1.3.4. Weight

Weight will be presented in kilograms. Weights reported in pounds will be converted as follows:

Weight in kilograms = Weight in pounds / 2.2

## 10.1.3.5. Height

Height will be presented in centimeters. Heights reported in feet and inches will be converted as follows:

Height in centimeters = Height in inches x = 2.54

#### 10.1.3.6. Body mass index (BMI)

BMI will be calculated as follows:

BMI = (Weight in kilograms) / (Height in meters) $^2$ 

## 10.1.3.7. Temperature

Temperatures will be presented in degrees Celsius (°C). Temperatures reported in degrees Fahrenheit (°F) will be converted as follows:

Temperature (Celsius) =  $((Temperature (Fahrenheit) - 32) \times 5)/9$ 

# 10.1.3.8. Numerical serology results

Numerical serology results will be derived from the content of IS.ISORRES in the SDTM dataset. For assays with a specific cut-off, the following derivation rules apply:

| IS.ISORRES | Derived value |
|---|---|
| "value" and value is >= cut-off | value |
| "value" and value is < cut-off | cut-off/2 |
| "value" and value is >ULOQ (applicable for RSV neutralizing assay) | ULOQ |
| "value" and value is <lloq (applicable="" assay)<="" for="" neutralizing="" rsv="" td=""><td>LLOQ/2</td></lloq> | LLOQ/2 |
| value" and value is >=LLOQ and <uloq (applicable="" assay)<="" for="" neutralizing="" rsv="" td=""><td>value</td></uloq> | value |
| All other cases | missing |

### 10.1.3.9. Geometric mean titers (GMTs) and concentrations (GMCs)

Geometric Mean Titer (GMT) or Concentration (GMC) calculations are performed by taking the inverse logarithm of the mean of the log titer or concentration transformations. Antibody titers or concentrations below the cut-off of the assay will be given an arbitrary value of half the cut-off of the assay for the purpose of GMT/GMC calculation. The cut-off value is defined by the laboratory before the analysis and is described in the protocol.

#### 10.1.3.10. Onset day

The onset day for an event (e.g. AE, medication, vaccination) is the number of days between the last study vaccination and the start date of the event. This is 1 for an event occurring on the same day as a vaccination (and reported as starting after vaccination).

#### 10.1.3.11. Duration of events

The duration of an event with a start and end date will be the number of days between the start and end dates plus one day, i.e. an event that starts on 03MAR2018 and ends on 12MAR2018 has a duration of 10 days.

The duration of solicited events will be calculated as the sum of the individual days with the symptom reported at grade 1 or higher.

## 10.1.3.12. Counting rules for combining solicited and unsolicited adverse events

For output combining solicited and unsolicited adverse events, all serious adverse events will be considered general events since the administration site flag is not included in the expedited adverse event CRF pages.

Multiple events with the same preferred term which start on the same day are counted as only one occurrence.

#### 10.1.3.13. Counting rules for occurrences of solicited adverse events

When the occurrences of solicited adverse events are summarized, each event recorded as having occurred during a specific period will be counted as only one occurrence regardless of the number of days on which it occurs. Also, in the case of co-administered study vaccines, an injection site reaction recorded for a subject following multiple vaccines will be counted as only one occurrence.

### 10.1.3.14. Display of decimals

## 10.1.3.15. Percentages

Percentages and their corresponding confidence limits will be displayed with:

- no decimals when there are fewer than 50 subjects in each tabulated group
- one decimal when there are at least 50 subjects in at least one tabulated group
  - Exceptions will be made for percentages that are not 0% or 100% but appear as 0% or 100% due to rounding. For these specific cases the number of decimals will be increased until the displayed value is no longer 0% or 100%. Examples are given in the following table.

| n/N | Displayed percentage |
|-------------|----------------------|
| 10/45 | 22% |
| 1/45 | 2% |
| 10/55 | 18.2% |
| 1/55 | 1.8% |
| 1/300 | 0.3% |
| 1/3000 | 0.03% |
| 1/30000 | 0.003% |
| 299/300 | 99.7% |
| 2999/3000 | 99.97% |
| 29999/30000 | 99.997% |

- The display of additional decimals for values close to 0% or 100% will be applied only to point estimates and not confidence limits, which can be rounded and displayed as 0% or 100%.
- Values of exactly 0% or 100% will be presented with no decimals regardless of the number of subjects per tabulated group.

#### 10.1.3.16. Differences in percentages

Differences in percentages and their corresponding confidence limits will be displayed with one more decimal than the maximum number used to display the individual percentages, for example the difference between two percentages displayed with one decimal will be displayed with two decimals.

## 10.1.3.17. Demographic/baseline characteristics statistics

The mean, median, and standard deviation for continuous baseline characteristics (height, weight, body mass index (BMI), pre-vaccination body temperature) will be presented with one decimal.

The minimum and maximum values and quartile values (if required) will be presented with the same number of decimals as the observed values.

The maxima and minima of transformed height variables will be displayed with no decimals.

The maxima and minima of transformed weight variables will be displayed with no decimals with the exception of values are below 10kg where one decimal will be displayed.

The maximum and minima of transformed body temperatures will be displayed with one decimal

#### 10.1.3.18. Serological summary statistics

The number of decimals used when displaying geometric mean titers (GMT) or concentrations (GMC) and their confidence limits is shown in the following table:

| <b>GMT or GMC value</b> | Number of decimals to display |
|-------------------------|-------------------------------|
| <0.1 | 3 |
| >=0.1 and $<10$ | 2 |
| >=10 and <1000 | 1 |
| >=1000 | 0 |

When multiple categories of GMT or GMC values are present in the same table, the number of decimals displayed should match that of the smallest category (i.e. the one with the higher number of decimals). For example, if GMT or GMC values of <0.1 appear in the same table as values of >=0.1 and <10, 3 decimals should be displayed for both

GMT or GMC ratios and their confidence limits will be displayed with 2 decimals regardless of the actual values.

#### 10.1.3.19. Statistical methodology

# 10.1.3.20. Exact confidence intervals around proportions

The exact confidence intervals around within-group proportions are derived using the method of Clopper and Pearson [Clopper, 1934].

# 10.1.3.21. Standardized asymptotic confidence intervals around differences in proportions

The standardized asymptotic confidence intervals around differences in proportions are derived using the method of Mietinnen and Nurminen [Miettinen, 1985].

204894 (RSV-PED-011) Statistical Analysis Plan Final

## 10.2. TFL and/or TFL ToC

The TFL ToC can be found in eTMF folder section 11.1.1. As the process of TFL came when the SAP was already developed using previous process, no separate TFL has been prepared. The mock template are present in the SAP in Section 13 and tables to be generated for synopsis, in-text, post-text and posting has been flagged in the TFL ToC for different timepoints when the analysis is planned.

204894 (RSV-PED-011) Statistical Analysis Plan Final

# 11. REFERENCES

Clopper CJ, Pearson E. The Use of Confidence or Fiducial Limits Illustrated in the case of the Binomial. *Biometrika*. 1934;26:404-13.

Miettinen, O. S. and Nurminen, M. Comparative analysis of two rates. Statistics in Medicine, 1985;4,213-226.

Kim HW, Canchola JG, Brandt CD, et al. Respiratory syncytial virus disease in infants despite prior administration of antigenic inactivated vaccine. *Am J Epidemiol*. 1969; 89(4): 422-34

# 12. LIST OF LISTINGS FOR THE FINAL ANALYSIS

The following listings will be generated using the macros developed by DSCS

Appendix Table I.B – Demography

Appendix Table IBii - Vital signs

Appendix Table I.Cii - Reason for visit not done

Appendix Table I.D - General medical history - Physical examination

Appendix Table I.Eii – Screening conclusion

Appendix Table I.I - Reason for not administration of vaccine

Appendix Table II.Ai - Solicited local adverse events

Appendix Table II.B - Solicited general adverse events

Appendix Table II.Ci - Unsolicited adverse events within (30) days post-vaccination

Appendix Table II.Cii - Unsolicited adverse events after (30) days post-vaccination

Appendix Table II.Di - Concomitant medications

Appendix Table II.Dii - Concomitant vaccinations

Appendix Table IV.A – Haematology and Biochemistry

Appendix Table V.A - RTI Assessment, Surveillance / Asymptomatic visit and Worsening data

Randomisation list

## 13. MOCK TABLES

Template 1 Number of subjects by country and center - <RSV 1D, RSV 2D, Comparator/Placebo> groups (Exposed Set)

| | | | h group><br>XXXX | | ch group><br>N=XXXX | | otal<br>XXXX |
|---|---|---|---|---|---|---|---|
| Country | Center-Investigator Name | n | % | n | % | n | % |
| <each country=""></each> | <each center-investigator="" name=""></each> | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| | All | XXX | XX.X | XXX | XX.X | XXX | XX.X |

Short group label = long group label

N = total number of subjects

n = number of subjects in a given center or country

 $% = n/N \times 100$ 

Center = GSK Biologicals assigned center number

Template 2 Summary of study completion with reasons for withdrawal <RSV 1D, RSV 2D, Comparator/Placebo> <groups> < pooled RSV 1D, RSV 2D, Comparator/Placebo groups> (Exposed Set)

| | | <each group=""><br/>N=XXXX</each> | | otal><br>(XXX |
|---|---|---|---|---|
| | n | % | n | % |
| Completed the study | XXX | XX.X | XXX | XX.X |
| Withdrawn from the study | XXX | XX.X | XXX | XX.X |
| Primary reason for withdrawal | | | | |
| Adverse Event Requiring Expedited Reporting | XXX | XX.X | XXX | XX.X |
| Unsolicited Non-Serious Adverse Event | XXX | XX.X | XXX | XX.X |
| Solicited Adverse Event | XXX | XX.X | XXX | XX.X |
| Protocol Deviation | XXX | XX.X | XXX | XX.X |
| Withdrawal By Subject | XXX | XX.X | XXX | XX.X |
| Sponsor Study Termination | XXX | XX.X | XXX | XX.X |
| Lost To Follow-up | XXX | XX.X | XXX | XX.X |
| Migrated / Moved From The Study Area | XXX | XX.X | XXX | XX.X |
| Other | XXX | XX.X | XXX | XX.X |

Short group label = long group label

Completed = number of subjects who completed last study visit

Withdrawn = number of subjects who did not come for the last study visit

Template 3 Summary of visit attendance/phone contact completion <RSV 1D, RSV 2D, Comparator/Placebo> groups (Exposed Set)

| | | <group 1=""><br/>N=XXXX</group> | | <group 2=""><br/>N=XXXX</group> | | otal<br>XXXX |
|---|---|---|---|---|---|---|
| | n | % | n | % | n | % |
| Visit 1 (Day 1) | | | | | | |
| Attended | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| Did not attend yet | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| Withdrawal at visit or earlier | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| Did not attend | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| Visit X (Day Y) | | | | | | |
| Phone contact X (Day Y) | | | | | | |
| Completed | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| Did not complete yet | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| Withdrawal at visit or earlier | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| Did not complete | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| Phone contact X (Day Y) | | | | | | |
| Visit X (Day Y) | | | | | | |
| Last study contact (Day Y) | | | | | | |
| Completed | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| Did not complete yet | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| Withdrawal at visit or earlier | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| Did not complete | XXX | XX.X | XXX | XX.X | XXX | XX.X |

Short group label = long group label

N = Number of subjects in each group or in total

n/% = number / percentage of subjects in a given category

Template 4 Summary of important protocol deviations leading to elimination from any analyses <RSV 1D, RSV 2D, Comparator/Placebo> <groups>< -pooled RSV 1D, RSV 2D, Comparator/Placebo groups>

| Category | | <each grou<="" th=""><th>ıb&gt;</th><th></th><th>Total</th><th></th></each> | ıb> | | Total | |
|---|---|---|---|---|---|---|
| Sub-category | | N=XXXX | | | N=XXXX | |
| | осс | n | % | осс | n | % |
| At least one important protocol | XXX | XXX | XX.X | XXX | XXX | XX.X |
| deviation | | | | | | |
| | XXX | XXX | XX.X | XXX | XXX | XX.X |
| <category 1=""></category> | XXX | XXX | XX.X | XXX | XXX | XX.X |
| <sub-category 1=""></sub-category> | XXX | XXX | XX.X | XXX | XXX | XX.X |
| <sub-category 2=""></sub-category> | | | | | | |
| | XXX | XXX | XX.X | XXX | XXX | XX.X |
| <category 2=""></category> | | | | | | |

Short group label = long group label

N = Total number of subjects

Occ = number of occurrences = number of important protocol deviations

n/% = number / percentage of subjects with important protocol deviations

Template 5 Summary of subject disposition from enrolled set to randomized set (Exposed Set)

| | Tot<br>N=X | |
|-----------------------------------------------|------------|------|
| | n | % |
| Withdrawals prior to randomization | XXX | XX.X |
| <withdrawal 1="" reason=""></withdrawal> | XXX | XX.X |
| <withdrawal 2="" reason=""></withdrawal> | XXX | XX.X |
| | XXX | XX.X |
| Number of subjects included in randomized set | XXX | XX.X |

Short group label = long group label

N = Number of subjects

n = number of subjects enrolled by center

% = n / Number of subjects with available results x 100

Summary of subject disposition from randomized set to exposed set Template 6

| | <group 1=""><br/>N=XXX</group> | | <group 2=""><br/>N=XXX</group> | | Tota | al |
|---|---|---|---|---|---|---|
| | | | | | N=XXX | |
| | N | % | N | % | N | % |
| Withdrawals | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| <withdrawal 1="" reason=""></withdrawal> | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| <withdrawal 2="" reason=""></withdrawal> | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| Eliminations | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| <elimination 1<="" reason="" td=""><td>XXX</td><td>XX.X</td><td>XXX</td><td>XX.X</td><td>XXX</td><td>XX.X</td></elimination> | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| (code)> <elimination 2<="" reason="" td=""><td>XXX</td><td>XX.X</td><td>XXX</td><td>XX.X</td><td>XXX</td><td>XX.X</td></elimination> | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| (code)> | XXX | XX.X | xxx | XX.X | XXX | XX.X |
| Number of subjects included in Exposed Set | | | | | | |

Short group label = long group label

N = Number of subjects

n = number of subjects enrolled by center

% = n / Number of subjects with available results x 100

Summary of subject disposition from Exposed Set to Per Protocol Template 7 Set at <Day 31/Day 61/end of first RSV season> <RSV 1D, RSV 2D, Comparator/Placebo> groups (Exposed set)

| | | oup 1> | | up 2> | Tota | |
|---|---|---|---|---|---|---|
| | N=XXX | | N= | XXX | N=XXX | |
| | n | % | n | % | n | % |
| Withdrawals | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| <withdrawal 1="" reason=""></withdrawal> | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| <withdrawal 2="" reason=""></withdrawal> | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| Eliminations | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| <elimination 1<="" reason="" td=""><td>XXX</td><td>XX.X</td><td>XXX</td><td>XX.X</td><td>XXX</td><td>XX.X</td></elimination> | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| (code)> | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| <elimination (code)="" 2="" reason=""></elimination> | | | | | | |
| | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| Number of subjects included in Per Protocol Set at <day 31="" 61="" day="" end="" first="" of="" rsv="" season=""></day> | | | | | | |

Short group label = long group label

N = Number of subjects

n = number of subjects enrolled by center

% = n / Number of subjects with available results x 100

204894 (RSV-PED-011) Statistical Analysis Plan Final

Summary of subject disposition from Exposed Set to End of study <RSV 1D, RSV 2D, Comparator/Placebo> groups (Exposed set) Template 8

| | <group 1=""><br/>N=XXX</group> | | <group 2=""><br/>N=XXX</group> | | Total<br>N=XXX | |
|---|---|---|---|---|---|---|
| | n | % | n | % | N | % |
| Eliminations | XXX | XX.X | XXX | XX.X | xxx | XX.X |
| <elimination 1<="" reason="" td=""><td>XXX</td><td>XX.X</td><td>XXX</td><td>XX.X</td><td>XXX</td><td>XX.X</td></elimination> | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| (code)><br><elimination 2<br="" reason="">(code)&gt;</elimination> | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| Withdrawals | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| <withdrawal 1="" reason=""> <withdrawal 2="" reason=""></withdrawal></withdrawal> | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| Number of subjects who | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| completed the study | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| Completed with 1 dose<br>Completed with X doses | XXX | XX.X | XXX | XX.X | XXX | XX.X |

Short group label = long group label

N = Number of subjects

n = number of subjects enrolled by center % = n / Number of subjects with available results x 100

Template 9 Deviations from protocol for age and intervals between study visits <RSV 1D, RSV 2D, Comparator/Placebo> groups (Exposed Set)

| Type of interval | Interval range | | | <grou< th=""><th>p 1&gt;</th><th><gr< th=""><th>oup 2</th><th></th></gr<></th></grou<> | p 1> | <gr< th=""><th>oup 2</th><th></th></gr<> | oup 2 |
|---|---|---|---|---|---|---|---|
| | | | | Value | % | Value | % |
| Age (years) at firs | t From <x> to <y></y></x> | N | | XXX | | XXX | |
| vaccine | years | n | | XXX | | XXX | XX.X |
| administration | | Below | XX.X | | | XXX | XX.X |
| | | <x></x> | | XXX | | XXX | XX.X |
| | | Above | XX.X | | | | |
| | | <y></y> | | XXX | | | |
| Number of days between vaccination <x> and vaccination <y></y></x> | From <x> to <y> days</y></x> | | XX.X | | | | |
| Number of days between vaccination <x></x> | From <x> to <y> days</y></x> | | | | | | |
| and visit <y></y> | From <x> to <y> days</y></x> | | | | | | |
| Number of days between vaccination <x> and blood sampling <y></y></x> | | | | | | | |

Short group label = long group label

N = total number of subjects with available results

n/% = number / percentage of subjects with results outside of the interval range = minimum-maximum for age and intervals

Template 10 Minimum and maximum visit dates <RSV 1D, RSV 2D, Comparator/Placebo> groups (Exposed Set)

| Visit Description | Parameter | <each group=""><br/>Date</each> | <each group=""><br/>Date</each> | Overall<br>Date |
|---|---|---|---|---|
| < each informed consent> | Minimum | DDMMYYYY | DDMMYYYY | DDMMYYYY |
| | Maximum | DDMMYYYY | DDMMYYYY | DDMMYYYY |
| [Randomization] | Minimum | DDMMYYYY | DDMMYYYY | DDMMYYYY |
| • | Maximum | DDMMYYYY | DDMMYYYY | DDMMYYYY |
| <each visit=""></each> | Minimum | DDMMYYYY | DDMMYYYY | DDMMYYYY |
| | Maximum | DDMMYYYY | DDMMYYYY | DDMMYYYY |
| Short group label = long group | label | | | |

204894 (RSV-PED-011) Statistical Analysis Plan Final

Template 11 Summary of demographic characteristics - <RSV 1D, RSV 2D, Comparator/Placebo> <groups>< -pooled RSV 1D, RSV 2D, Comparator/Placebo groups> (Exposed Set, PPS for immunogenicity at <Day 31/Day 61/end of first RSV season>)

| <group 1<="" th=""><th><b> </b>&gt;</th><th><group 2=""></group></th><th>&gt;</th><th><group 3<="" th=""><th>&gt;</th><th>Total</th><th></th></group></th></group> | <b> </b> > | <group 2=""></group> | > | <group 3<="" th=""><th>&gt;</th><th>Total</th><th></th></group> | > | Total | |
|---|---|---|---|---|---|---|---|
| N = | | N = | | N = | | N = | |
| Value or n | % | Value or n | % | Value or n | % | Value or n | % |

Age (months) at first vaccination

n

Mean

Standard Deviation

Median

Minimum

Maximum

Sex

Female

Male

Geographic Ancestry

African Heritage / African American

American Indian or Alaskan Native

Asian - Central/South Asian Heritage

Asian - East Asian Heritage

Asian - Japanese Heritage

Asian - South East Asian Heritage

Native Hawaiian or Other Pacific Islander

White - Arabic / North African Heritage

White - Caucasian / European Heritage

Other

#### <each group>:

N = total number of subjects

n/% = number / percentage of subjects in a given category

Value = value of the considered parameter

SD = standard deviation

204894 (RSV-PED-011) Statistical Analysis Plan Final

Template 12 Summary of vital signs characteristics - <RSV 1D, RSV 2D,
Comparator/Placebo> <groups>< pooled RSV 1D, RSV 2D,
Comparator/Placebo groups> (Exposed set, PPS for immunogenicity at <Day 31/Day 61/end of first RSV season>)

| | | | <each group=""><br/>N =</each> | Total<br>N = |
|---|---|---|---|---|
| Visit | Characteristics | Parameters | Value | Value |
| <each visit=""></each> | Height (Cm) | N with data | | |
| | | Mean | | |
| | | SD | | |
| | | Median | | |
| | | Minimum | | |
| | | Maximum | | |
| | Weight (Kg) | N with data | | |
| | | Mean | | |
| | | SD | | |
| | | Median | | |
| | | Minimum | | |
| | | Maximum | | |
| | Heart rate (Beats per minute) | N with data | | |
| | | Mean | | |
| | | SD | | |
| | | Median | | |
| | | Minimum | | |
| | | Maximum | | |
| | Respiratory rate (Breadth per minute) | N with data | | |
| | | Mean | | |
| | | SD | | |
| | | Median | | |
| | | Minimum | | |
| | | Maximum | | |
| | Temperature/(Axillary) (°C) | N with data | | |
| | | Mean | | |
| | | SD | | |
| | | Median | | |
| | | Minimum | | |
| | | Maximum | | |

#### <each group>:

N = total number of subjects

N with data = number of subjects with documentation of the corresponding data

Value = value of the considered parameter

SD = standard deviation

Template 13 Number of enrolled subjects by age category <RSV 1D, RSV 2D, Comparator/Placebo> groups

| | | <each group=""><br/>N =</each> | Total<br>N = |
|---|---|---|---|
| Characteristics | Categories | n | n |
| Age category | 1=Infants and toddlers (28 days-23 month) Missing | | |

#### <each group>:

N = Number of enrolled subjects

n= number of enrolled subjects included in each group or in total for a given age category or for all age categories Missing = age at dose 1 unknown

Template 14 Compliance in completing solicited adverse events information <RSV 1D, RSV 2D, Comparator/Placebo> groups (Exposed Set)

| | | <group 1=""></group> | | | | <group< th=""><th>2&gt;</th></group<> | 2> |
|---|---|---|---|---|---|---|---|
| | | N | n | | N | n | |
| | | Compliand | e | | Complia | nce | |
| | | | | (%) | | | (%) |
| < Vaccination at vi | sit General solicited adverse | XXX | XXX | XX.X | XXX | XXX | XX.X |
| 1> | events | XXX | XXX | XX.X | XXX | XXX | XX.X |
| | Local solicited adverse events | | | | | | |
| <vaccination at="" td="" vi<=""><td>sit</td><td>XXX</td><td>XXX</td><td>XX.X</td><td>XXX</td><td>XXX</td><td>XX.X</td></vaccination> | sit | XXX | XXX | XX.X | XXX | XXX | XX.X |
| X> | General solicited adverse events | XXX | XXX | XX.X | XXX | XXX | XX.X |
| Per vaccination | Local solicited adverse events | XXX | | XX.X | XXX | XXX | XX.X |
| | | XXX | | XX.X | XXX | XXX | XX.X |
| | General solicited adverse events | XXX | XXX | | | | |
| | Local solicited adverse events | | | | | | |

Short group label = long group label

N=Number of administered vaccination

n = number of vaccination with Adverse Event Screen returned

Compliance (%) =  $(n / N) \times 100$ 

204894 (RSV-PED-011) Statistical Analysis Plan Final

Template 15 Summary of <grade 3> adverse events (solicited and unsolicited)
<with causal relationship to vaccination, with medically attend visit>
within <7, 30> days following first and second vaccination and
overall <RSV 1D, RSV 2D, Comparator/Placebo> <groups>< pooled
RSV 1D, RSV 2D, Comparator/Placebo groups> (Exposed Set)

| | | <each group=""></each> | | | |
|---|---|---|---|---|---|
| | | | | 95 | % CI |
| | | n | % | LL | UL |
| <vaccination 1="" at="" visit=""></vaccination> | N | XXX | | | |
| | Any adverse event | XXX | XX.X | XX.X | XX.X |
| | Local adverse event | XXX | XX.X | XX.X | XX.X |
| | General adverse event | XXX | XX.X | XX.X | XX.X |
| <vaccination at="" visit="" x=""></vaccination> | | | | | |

Per subject

Per vaccination

Short group label = long group label

For each vaccination:

N = number of subjects with the corresponding administered vaccination

n/% = number/percentage of subjects presenting at least one type of adverse event following the corresponding dose For per vaccination:

N = number of administered vaccination

n/% = number/percentage of vaccination followed by at least one type of adverse event For per subject:

N = number of subjects with at least one administered vaccination

n/% = number/percentage of subjects presenting at least one type of adverse event

95% CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

204894 (RSV-PED-011) Statistical Analysis Plan Final

Template 16 Percentage of subjects with solicited local adverse events by maximum intensity within the 7-day (Days 1-7) following first and second vaccination and overall - <RSV 1D, RSV 2D, Comparator/Placebo> <groups> < pooled RSV 1D, RSV 2D, Comparator/Placebo groups>(Exposed Set)

Adverse event: Pain

| | | <group 1=""></group> | | | | | <gro< th=""><th colspan="4">oup 2&gt;</th></gro<> | oup 2> | |
|---|---|---|---|---|---|---|---|---|---|
| | | 95% CI | | | | 95% CI | | | |
| | | n | % | LL | UL | n | % | LL | UL |
| <pre><vaccination 1="" at="" visit=""></vaccination></pre> | N | XXX | | | | XXX | | | |
| | Any | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| | Grade 2 | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| | Grade 3 | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| | Medically attended visits | | | | | | | | |

<sup>&</sup>lt;Vaccination at visit 3>

Per subject

Per vaccination

Adverse event: Swelling/Redness

| | | <group 1=""></group> | | | | | <gro< th=""><th colspan="4">Group 2&gt;</th></gro<> | Group 2> | |
|---|---|---|---|---|---|---|---|---|---|
| | | 95% CI | | | | 95% CI | | | |
| | | n | % | LL | UL | n | % | LL | UL |
| <vaccination 1="" at="" visit=""></vaccination> | N | XXX | | | | XXX | | | |
| | Any | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| | ≥5 - ≤ 20 | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| | >20 | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| | Medically attended visits | | | | | | | | |

<sup>&</sup>lt;Vaccination at visit 3>

Per subject

Per vaccination

#### <each group>:

For each vaccination:

N = number of subjects with the corresponding documented vaccination

n/% = number/percentage of subjects reporting the type of adverse event at least once following the corresponding vaccination

For Per vaccination:

N = number of documented vaccination

n/% = number/percentage of vaccination followed by at least one type of adverse event

For Per subject:

N = number of subjects with at least one documented vaccination

204894 (RSV-PED-011) Statistical Analysis Plan Final

n/% = number/percentage of subjects reporting the type of adverse event at least once 95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

The maximum intensity of local injection site redness/swelling was coded as follows:

- 1: > 0.1 mm to < 5 mm
- $2: \geq 5 \text{ mm to} \leq 20 \text{ mm}$
- 3: > 20 mm

Please note – The N may vary for each symptom depending on how many subjects has filled in diary card for particular symptom.

Template 17 Duration in days of solicited <general, local> adverse events within 7 days following first and second vaccination and overall <RSV 1D, RSV 2D, Comparator/Placebo> groups (Exposed Set)

| | Symptom | <group 1=""></group> | <group 2=""></group> |
|---|---|---|---|
| | | Value | Value |
| <vaccination at<="" td=""><td><symptom 1=""></symptom></td><td></td><td></td></vaccination> | <symptom 1=""></symptom> | | |
| visit 1> | n | xxx | XXX |
| | Mean | XXX.X | XXX.X |
| | Minimum | XXX | XXX |
| | Q1 | XXX.X | XXX.X |
| | Median | XXX.X | XXX.X |
| | Q3 | XXX.X | XXX.X |
| | Maximum | XXX | XXX |

<Vaccination at visit X>

#### Per vaccination

Short group label = long group label

n = number of doses with the adverse event

<Symptom 2>

Q1 = 25th percentile

Q3 = 75th percentile

204894 (RSV-PED-011) Statistical Analysis Plan Final

Template 18 Percentage of subjects with solicited general adverse events by maximum intensity within the 7-day (Days 1-7) following first and second vaccination and overall - <RSV 1D, RSV 2D, Comparator/Placebo> <groups> < pooled RSV 1D, RSV 2D, Comparator/Placebo groups > (Exposed Set)

Adverse event: Irritability/Fussiness or Drowsiness or Loss of appetite

| | | <group 1=""></group> | | | | | <group 2=""></group> | | |
|---|---|---|---|---|---|---|---|---|---|
| | | 95% CI | | | | | 95% C | | |
| | | n | % | LL | UL | n | % | LL | UL |
| <vaccination 1="" at="" visit=""></vaccination> | N | XXX | | | | XXX | | | |
| | Any | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| | Grade 2 | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| | Grade 3 | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| | Any related | | | | | | | | |
| | Grade 2 related | | | | | | | | |
| | Grade 3 related | | | | | | | | |
| | Medically attended visits | | | | | | | | |
| diametra | • | | | | | | | | |

<Vaccination at visit 3>

Per subject

Per vaccination

Adverse event: Temperature (C)

| | | <group 1=""></group> | | | | | <group 2=""></group> | | |
|---|---|---|---|---|---|---|---|---|---|
| | | 95% CI | | | | | 95% CI | | |
| | | n | % | LL | UL | n | % | LL | UL |
| <vaccination 1="" at="" visit=""></vaccination> | N | XXX | | | | XXX | | | |
| | Any | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| | ≥38.0 | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| | ≥38.5 | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| | ≥39.0 | | | | | | | | |
| | ≥39.5 | | | | | | | | |
| | >40.0 | | | | | | | | |
| | Related | | | | | | | | |
| | >39.0 - ≤40.0 Related | | | | | | | | |
| | >40.0 Related | | | | | | | | |
| | Medically attended visits | | | | | | | | |

<Vaccination at visit 3>

Per subject Per vaccination

#### <each group>:

For each vaccination:

N = number of subjects with the corresponding documented vaccination

n/% = number/percentage of subjects reporting the type of adverse event at least once following the corresponding vaccination

For Per vaccination:

N = number of documented vaccination

n/% = number/percentage of vaccination followed by at least one type of adverse event

For Per subject:

N = number of subjects with at least one documented vaccination

n/% = number/percentage of subjects reporting the type of adverse event at least once

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

Please note – The N may vary for each adverse event depending on how many subjects has filled in diary card for particular symptom.

Template 19 Percentage of subjects reporting solicited local adverse events (any grade /grade 2,3/ grade 3) within 7-days following first and second vaccination by maximum intensity for pooled RSV 1D, RSV 2D, Comparator/Placebo groups (Exposed Set)



<each group>

Please note - this graph will be presented on pooled group only

Template 20 Percentage of subjects reporting fever (any and grade 3) and other solicited general adverse events (any grade /grade 2,3/ grade 3) within 7-days following first and second vaccination by maximum intensity for pooled RSV 1D, RSV 2D and Comparator/Placebo groups (Exposed Set)



<each group>

Please note the figure is only template

Please note – this graph will be presented on pooled group only

Template 21 Summary of subjects with at least one <Ø/grade 3/ related/ grade 3 related/serious/ medically attended> unsolicited adverse event <episode of spontaneous or excessive bleeding> classified by MedDRA Primary System Organ Class and Preferred Term <with onset within 30 days of first and second vaccination><from vaccination dose 1 up to Day 61> <pooled> <RSV 1D, RSV 2D, Comparator/Placebo> groups (Exposed Set)

| | | | up 1> | | <group 2=""><br/>N=XXXX</group> | | | |
|---|---|---|---|---|---|---|---|---|
| Primary System Organ Class (CODE) | | | 95 | | % CI | | | |
| Preferred Term (CODE) | n | % | LL | UL | N | % | LL | UL |
| Any <Ø, grade 3, related, grade3 related> unsolicited adverse event | XXX | XX.X | XX.X | XX.X | Xxx | XX.X | XX.X | XX.X |
| <soc (code)="" 1=""></soc> | XXX | XX.X | XX.X | XX.X | Xxx | XX.X | XX.X | XX.X |
| <preferred (code)="" 1="" term=""></preferred> | XXX | XX.X | XX.X | XX.X | Xxx | XX.X | XX.X | XX.X |
| <pre><pre>referred Term 2 (code)&gt;</pre></pre> | XXX | XX.X | XX.X | XX.X | Xxx | XX.X | XX.X | XX.X |
| <soc (code)="" 2=""></soc> | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| <pre><pre>referred Term 1 (code)&gt;</pre></pre> | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| <preferred (code)="" 2="" term=""></preferred> | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |

Short group label = long group label

Any adverse event = at least one adverse event experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with at least one administered vaccination

n\* = number of events reported

n/% = number/percentage of subjects reporting the adverse event at least once

<sup>95%</sup> CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Template 22 Summary of subjects with at least one <episode of RSV-LRTI (AE of specific interest)/serious adverse event> classified by MedDRA Primary System Organ Class and Preferred Term <from vaccination dose 1 up to end of <first/second> RSV season for pooled RSV 1D, RSV 2D and Comparator/Placebo groups (Exposed Set)

| | <group 1=""></group> | | | | <group 2=""></group> | | | |
|---|---|---|---|---|---|---|---|---|
| | | N=X | XXX | | N=XXXX | | | |
| Primary System Organ Class (CODE) | 95% CI | | | | | | 95% CI | |
| Preferred Term (CODE) | n | % | LL | UL | N | % | LL | UL |
| Any <Ø, grade 3, related, grade3 related> unsolicited adverse event | XXX | XX.X | XX.X | XX.X | Xxx | XX.X | XX.X | XX.X |
| <soc (code)="" 1=""></soc> | XXX | XX.X | XX.X | XX.X | Xxx | XX.X | XX.X | XX.X |
| <preferred (code)="" 1="" term=""></preferred> | XXX | XX.X | XX.X | XX.X | Xxx | XX.X | XX.X | XX.X |
| <pre><pre>referred Term 2 (code)&gt;</pre></pre> | XXX | XX.X | XX.X | XX.X | Xxx | XX.X | XX.X | XX.X |
| <soc (code)="" 2=""></soc> | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| <preferred (code)="" 1="" term=""></preferred> | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| <preferred (code)="" 2="" term=""></preferred> | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |

Short group label = long group label

Any adverse event = at least one adverse event experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with at least one administered vaccination

n\* = number of events reported

n/% = number/percentage of subjects reporting the adverse event at least once

<sup>95%</sup> CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit
204894 (RSV-PED-011) Statistical Analysis Plan Final

# Template 23 Listing of SAE from vaccination dose 1 up to <Day 61/end of first RSV season/study end> (Exposed Set)

| Group | Subject<br>number | Gender | Country | Race | Age at onset (Year) | Verba | tim | Preferr | ed Term |
|---|---|---|---|---|---|---|---|---|---|
| XXXXX | xxxxx | xxxxx | XXXXXXX | XXXXXX | xx | xxxxx | | xxxxx | |
| Group | - | Primary Syste<br>Organ Class | m Medical<br>visit type | Vaccin<br>ation | Day of onset | Duration | Intensity | Causality | Outco<br>me |
| xxxxx | xxxxx | xxxxx | xxxxxx | xxxxxx | XX | xx | xxxx | 1 | xxxxx |
| Group | Subject<br>number | Seriousness<br>criteria | Potential<br>AESI<br>(prefered<br>term) | | | | | <u> </u> | |
| xxxxx | XXXXX | xxxxx | xxxxxxx | xxxxx | xx | xx | xxxx | 1 | xxxxx |

Template 24 Listing of AEs related to LRTI and association to RSV infection from vaccination dose 1 up to <Day 61/end of first RSV season/study end> (Exposed Set)

| Gro | Su | Age | Verba | Prefer | ME | Previ | Day | Sta | En | Durati | Intens | Causa | Outco | Loc | Date | Cent | Cent | Date | ΑE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| up | b. | at | tim | red | D | ous | of | rt | d | on | ity | lity | me | al | of | ral | ral | of | SI |
| | No | onset | | term | typ | Dose | ons | dat | da | | | | | RS | sam | test | test | sam | |
| | | (mon | | | е | | et | е | te | | | | | ٧ | ple | RSV | RSV | ple | |
| | | th) | | | | | | | | | | | | test | for | Α | В | for | |
| | | | | | | | | | | | | | | res | local | | | centr | |
| | | | | | | | | | | | | | | ult | testi | | | al | |
| | | | | | | | | | | | | | | | ng | | | testi | |
| | | | | | | | | | | | | | | | | | | ng | |

<sup>&</sup>lt;each group>:

AESI: AEs of Special Interest - LRTI identified by the Investigator

<sup>\*</sup>AEs related to LRTI will be identified based on the list of preferred terms described in in section 9.4–Annex 2

Template 25 Listing of AEs related to spontaneous or excessive bleeding together with hemoglobin and platelet count results with 30 days of first and second vaccination (Exposed Set)

| Gr<br>ou<br>p | Sub. | Age<br>at<br>ons<br>et<br>(mo<br>nth) | Verb<br>atim | Preferre d term* | Prev<br>ious<br>Dos<br>e | Da<br>y<br>of<br>on<br>set | Dura<br>tion | Inte<br>nsit<br>y | Start<br>date | End<br>date | A<br>E<br>SI | Dat<br>e of<br>sa<br>mpl<br>e | Labor<br>atory<br>param<br>eter | Ra<br>w<br>res<br>ult | U<br>ni<br>t |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XX | | | | | | XX | | | | | | | Hemo | | |
| | XX | | XX | XX | XX | | | | XX | XX | | XX | globin | | |
| | | | | | | | | | | | | | Platel | | |
| | | | | | | | | | | | | | et | | |
| | | | | | | | | | | | | | count | | |
| | | | | | | | | | | | | | Hemo | | |
| | | | | | | | | | | | | XX | globin | | |
| | | | | | | | | | | | | | Platel | | |
| | | | | | | | | | | | | | et | | |
| | | | | | | | | | | | | | count | | |

<sup>&</sup>lt;each group>:

AESI: AEs of Special Interest - Spontaneous or excessive bleeding identified by the Investigator

Template 26 Listing of adverse events, SAEs and solicited symptoms leading to study or treatment discontinuation from vaccination dose 1 up to <Day 61/end of first RSV season/end of second RSV season>(Exposed Set)

Type of discontinuation: <study/treatment>

| Group | Subject<br>number | Gender | Country | Race | AE<br>Description | SAE (Y/N) | Causalit | y Outcome | Vaccination and visit |
|---|---|---|---|---|---|---|---|---|---|
| XXXXX | XXXXX | XXXXX | XXXXXXX | XXXXXX | XXXXXX | Х | XXXXX<br>X | XXXXX | Vaccination: x at visit |

## Template 27 Listing of unscheduled safety visit from vaccination dose 1 up to <Day 61/end of first RSV season/study end> (Exposed Set)

| Group | Sub.No. | Cou<br>ntry | unschedul<br>ed visit | previous | unscheduled | safety<br>BS out of | abnormality<br>per protocol –<br>previous | biochemistry/<br>hematology at |
|---|---|---|---|---|---|---|---|---|

#### <each group>:

Please note that only unscheduled safety visits with abnormal safety parameters will be presented.

<sup>\*</sup>AEs related to spontaneous or excessive bleeding will be identified based on the list of preferred terms described in section 9.4 –Annex

204894 (RSV-PED-011) Statistical Analysis Plan Final

Template 28 Summary of subjects taking a concomitant medication within <7/30>
days following each vaccination and overall <RSV 1D, RSV 2D,
Comparator/Placebo> <groups>< for pooled RSV 1D, RSV 2D and
Comparator/Placebo groups> (Exposed Set)

| | | | <gro< th=""><th>up 1&gt;</th><th></th><th colspan="6"><group 2=""></group></th></gro<> | up 1> | | <group 2=""></group> | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | 95% CI 95% CI | | | | | | | |
| | | n | % | LL | UL | n | % | LL | UL |
| <vaccination 1="" at="" visit=""></vaccination> | N | XXX | | | | XXX | | | |
| | Any | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| | Any antipyretic | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| | Any prophylactic antipyretic | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |

<Vaccination at visit X>

Per subject

## Per vaccination

Short group label = long group label

For each vaccination:

N = number of subjects with the corresponding administered vaccination

n/% = number/percentage of subjects who took the specified type of concomitant medication at least once during the considered period

For per vaccination:

N = number of administered vaccination

n/% = number/percentage of vaccines after which the specified type of concomitant medication was taken at least once during the considered period

For per subject:

N = number of subjects with at least one administered vaccination

n/% = number/percentage of subjects who took the specified type of concomitant medication at least once during the considered period

95% CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

Template 29 Summary of occurrences and subjects with at least one solicited and unsolicited adverse event classified by MedDRA Primary System Organ Class and Preferred Term with onset within 30 days of first and second vaccination – SAE excluded <RSV 1D, RSV 2D, Comparator/Placebo> groups (Exposed Set)

| Primary System Organ Class (CODE) | | Group 1<br>N=XXXX | | | <group 2=""><br/>N=XXXX</group> | • |
|---|---|---|---|---|---|---|
| Preferred Term (CODE) | осс | n | % | осс | n | % |
| Any solicited and unsolicited adverse event | XXX | xxx | XX.X | XXX | xxx | XX.X |
| <soc (code)="" 1=""></soc> | XXX | XXX | XX.X | XXX | XXX | XX.X |
| <preferred (code)="" 1="" term=""></preferred> | XXX | XXX | XX.X | XXX | XXX | XX.X |
| <pre><preferred (code)="" 2="" term=""></preferred></pre> | XXX | XXX | XX.X | XXX | XXX | XX.X |
| <soc (code)="" 2=""></soc> | XXX | XXX | XX.X | xxx | XXX | XX.X |
| <preferred (code)="" 1="" term=""></preferred> | XXX | XXX | XX.X | XXX | XXX | XX.X |
| <preferred (code)="" 2="" term=""></preferred> | XXX | XXX | XX.X | XXX | XXX | XX.X |

Short group label = long group label

Any adverse event = at least one adverse event experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with at least one administered vaccination

n\* = number of events reported

n/% = number/percentage of subjects reporting the adverse event at least once

<sup>95%</sup> CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

204894 (RSV-PED-011) Statistical Analysis Plan Final

Template 30 Number (%) of subjects with serious adverse events <from Day 1 up to <Day 61/end of second RSV season>, including number of events reported for pooled RSV 1D, RSV 2D and Comparator/Placebo> groups (Exposed Set)

| | | | <eacl< th=""><th>h group</th><th>&gt;</th><th><eacl< th=""><th>n group&gt;<br/>XX</th><th>•</th></eacl<></th></eacl<> | h group | > | <eacl< th=""><th>n group&gt;<br/>XX</th><th>•</th></eacl<> | n group><br>XX | • |
|---|---|---|---|---|---|---|---|---|
| Type of Event | Primary System Organ Class (CODE) | Preferred Term<br>(CODE) | n* | n | % | n* | n | % |
| SAE | | At least one symptom | XXX | XXX | XX.X | XXX | XXX | XX.X |
| | <pre><each (soc="" code)="" soc=""></each></pre> | <each (pt="" code)="" pt=""></each> | XXX | XXX | XX.X | XXX | XXX | XX.X |
| ı | | At least one symptom | | XXX | XX.X | XXX | XXX | XX.X |
| Related SAE | | At least one symptom | XXX | XXX | XX.X | XXX | XXX | XX.X |
| Neialeu SAL | <pre><each (soc="" code)="" soc=""></each></pre> | <each (pt="" code)="" pt=""></each> | XXX | XXX | XX.X | XXX | XXX | XX.X |
| | | | XXX | XXX | XX.X | XXX | XXX | XX.X |
| Fatal SAE | | At least one symptom | xxx | XXX | XX.X | XXX | XXX | XX.X |
| | <each (soc="" code)="" soc=""></each> | <each (pt="" code)="" pt=""></each> | xxx | XXX | XX.X | XXX | XXX | XX.X |
| | | | XXX | XXX | XX.X | XXX | XXX | XX.X |
| Related Fatal | | At least one symptom | XXX | XXX | XX.X | XXX | XXX | XX.X |
| SAE | <each (soc="" code)="" soc=""></each> | <each (pt="" code)="" pt=""></each> | xxx | XXX | XX.X | XXX | XXX | XX.X |
| | | | XXX | XXX | XX.X | XXX | XXX | XX.X |

Short group label = long group label

N = number of subjects with administered vaccination

n/% = number/percentage of subjects reporting the adverse event at least once

n\* = Number of adverse events reported

Related = assessed by the investigator as related

Template 31 Number and percentage of subjects with <anti-RSV A antibody titre, anti-RSV F concentration> equal to or above <cut-off ><unit> and gm<t,c> for pooled RSV 1D, RSV 2D and Comparator/Placebo> groups (<Adapted>PPS of immunogenicity at <Day X, end of 1st RSV season>)

| Antibody<br>off | Time point | Cut- | | | <grou< th=""><th>p 1&gt;</th><th></th><th></th><th>&lt;(</th><th>Group 2</th><th>2&gt;</th><th></th></grou<> | p 1> | | | <( | Group 2 | 2> | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 959 | % CI | | | | 959 | % CI |
| | | | N | n | value | LL | UL | N | n | value | LL | UL |
| <antibody 1=""> off 1&gt;</antibody> | 1> <time 1<="" point="" td=""><td>&gt; <cut-%>=<cut-off 1=""><br/><unit></unit></cut-off></cut-%></td><td>XXX</td><td>XXX</td><td>XX.X</td><td>XX.X</td><td>XX.X</td><td>XXX</td><td>XXX</td><td>XX.X</td><td>XX.X</td><td>XX.X</td></time> | > <cut-%>=<cut-off 1=""><br/><unit></unit></cut-off></cut-%> | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | | GM <t,c></t,c> | xxx | | XX.X | XX.X | XX.X | XXX | | XX.X | xx.x | |
| | | | | | | | | | | | | XX.X |

Short group label = long group label

GMT/C = geometric mean antibody titer/concentration

N = Number of subjects with available results

n/% = number/percentage of subjects with titer/concentration equal to or above specified value

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

PRE= Pre-vaccination

D31 = Post-vaccination at Day 31

D61 = Post-vaccination at Day 61

204894 (RSV-PED-011) Statistical Analysis Plan Final

Template 32 Distribution of <RSV-A neutralising antibody titre, RSV-F antibody concentration> for pooled RSV 1D, RSV 2D and Comparator/Placebo> groups (<Adapted>PPS for immunogenicity <at Day X, end of 1st RSV season>)

| Antibody | Time point | Cut-off | | | <group< th=""><th>1&gt;</th><th></th><th></th><th><g< th=""><th>roup 2&gt;</th><th>•</th><th></th></g<></th></group<> | 1> | | | <g< th=""><th>roup 2&gt;</th><th>•</th><th></th></g<> | roup 2> | • | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 95% | CI | | | | 95% | CI |
| | | | N | n | value | LL | UL | N | n | value | LL | UL |
| <antibody 1=""></antibody> | <time 1="" point=""></time> | <cut-off 1<="" td=""><td>XXX</td><td>XXX</td><td>XX.X</td><td>XX.X</td><td>XX.X</td><td>XXX</td><td>XXX</td><td>XX.X</td><td>XX.X</td><td>XX.X</td></cut-off> | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | | >=cut-off 2 | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | | >=cut-off 3 | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | <time 2="" point=""></time> | <cut-off 1<="" td=""><td>XXX</td><td>XXX</td><td>XX.X</td><td>XX.X</td><td>XX.X</td><td>XXX</td><td>XXX</td><td>XX.X</td><td>XX.X</td><td>XX.X</td></cut-off> | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | | >=cut-off 2 | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | | >=cut-off 3 | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |

Short group label = long group label

N = number of subjects with available results

n/% = number/percentage of subjects with <titer, concentration> within the specified criterion

<95>% CI = <95>% confidence interval; LL = Lower Limit, UL = Upper Limit

PRE= Pre-vaccination

D31 = Post-vaccination at Day 31

D61 = Post-vaccination at Day 61

Template 33 Vaccine response for anti-RSV-A neutralising antibody titre at each post-vaccination timepoint for pooled RSV 1D, RSV 2D and Comparator/Placebo> groups (PPS for analysis of immunogenicity at <Day X, End of 1st RSV season>)

| Antibody | Time point | Pre-vaccination | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Category | | | <gr< th=""><th>oup 1&gt;</th><th>•</th><th></th><th>&lt;</th><th>Group</th><th>2&gt;</th><th></th></gr<> | oup 1> | • | | < | Group | 2> | |
| | | | | | | 959 | % CI | | | | 9 | 5% CI |
| | | | N | n | value | LL | UL | N | n | value | LL | UL |
| <antibody 1=""></antibody> | > <time point<="" td=""><td>&lt;128</td><td>XXX</td><td>XXX</td><td>XX.X</td><td>XX.X</td><td>XX.X</td><td>XXX</td><td>XXX</td><td>XX.X</td><td>XX.X</td><td>XX.X</td></time> | <128 | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | | ≥128 - ≤256 | XXX | XXX | XX.X | XX.X | XX.X | XXX | xxx | XX.X | XX.X | XX.X |
| | | >256-≤1024 | XXX | XXX | XX.X | XX.X | XX.X | xxx | XXX | XX.X | XX.X | XX.X |
| | | ≥1024<br>Total response | XXX | XXX | XX.X | xx.x | XX.X | XXX | XXX | XX.X | XX.X | XX.X |

Short group label = long group label

Total = all subjects with pre-and post- vaccination result available

Vaccine response defined as:

For subjects with pre-vaccination titer <128: antibody titer at post-vaccination>= 4 fold the pre-vaccination antibody titer

For subjects with pre-vaccination titer in ≥128 - ≤256: antibody titer at post-vaccination >= 3 fold the pre-vaccination antibody titer

For subjects with pre-vaccination titer in >256-≤1024: antibody titer at post-vaccination>= 2.5 fold the pre-vaccination antibody titer

For subjects with pre-vaccination titer >1024: antibody titer at post-vaccination >= 1 fold the pre-vaccination antibody titer

N = number of subjects with both pre- and post-vaccination results available

n/% = number/percentage of responders

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

PRE= Pre-vaccination

<D31 = Post-vaccination at Day 31>

<D61 = Post-vaccination at Day 61>

204894 (RSV-PED-011) Statistical Analysis Plan Final

Template 34 Number and percentage of subjects with <anti-RSV A antibody titre, anti-RSV F concentration> equal to or above <cut-off ><unit> and GMR for pooled RSV 1D, RSV 2D and Comparator/Placebo> groups (PPS of immunogenicity at <Day X, End of 1st RSV season>)

| Antibody | Time point | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Cut-off | | | | | <grou< th=""><th>p 1&gt;</th><th></th><th></th><th></th><th><gro< th=""><th>up 2&gt;</th><th></th></gro<></th></grou<> | p 1> | | | | <gro< th=""><th>up 2&gt;</th><th></th></gro<> | up 2> | |
| | | | | | | 95% | CI | | | | 959 | % CI |
| | | | N | n | value | LL | UL | N | n | value | LL | UL |
| <antibody 1=""><br/><cut-off 1=""></cut-off></antibody> | <time 1="" point=""></time> | %>= <cut-off 1=""> <unit></unit></cut-off> | XXX | xxx | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | | GMC/T<br>Visit comparison /<br>baseline | XXX | | XX.X | XX.X | XX.X | XXX | | XX.X | XX.X | XX.X |
| | | GMR | XXX | | XX.X | XX.X | XX.X | XXX | | XX.X | XX.X | XX.X |

Short group label = long group label

GMT = geometric mean antibody titer

N = Number of subjects with available results at the two considered time points

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

PRE= Pre-vaccination

D31 = Post-vaccination at Day 31

D61 = Post-vaccination at Day 61

204894 (RSV-PED-011) Statistical Analysis Plan Final

Template 35 Distribution of fold of anti-RSV-A neutralising antibody titer by <cumulative> pre-vaccination titer category for pooled RSV 1D, RSV 2D and Comparator/Placebo> groups (PPS for analysis of immunogenicity at <Day X, end of first RSV season>)

| Antibody | Time point | Pre-vaccination | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Fold | • | status | | <0 | roup 1 | > | | | <( | roup | 2> | |
| | | | | | 95% ( | CI | | | 9 | 5% CI | | |
| | | | N | n | Value | LL | UL | N | n | Value | LL | UL |
| <antibody 1=""></antibody> | <time 1="" point=""> &lt;1</time> | <128 | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | | ≥128-≤256 | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | | >256-≤512 | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | | >1024-≤2048 | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | | >2048-≤4096 | | Ххх | XX.X | XX.X | xx.x | XXX | XXX | XX.X | XX.X | XX.X |
| | | | XXX | | | | | | | | | |
| | | >4096 | | Ххх | XX.X | XX.X | xx.x | XXX | XXX | XX.X | XX.X | XX.X |
| | | | XXX | | | | | | | | | |
| | | Total | | XXX | XX.X | XX.X | XX.X | XXX | ( XXX | XX.X | XX.X | XX.X |
| | | | XXX | | | | | | | | | |
| | ≥1 | <128 <unit></unit> | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | ≥2 | <128 <unit></unit> | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |

Short group label = long group label

N = number of subjects with pre and corresponding post-vaccination results available

n/% = number/percentage of subjects with titre fold change meeting the specified criterion

PRE= Pre-vaccination

D31 = Post-vaccination at Day 31

D61 = Post-vaccination at Day 61

204894 (RSV-PED-011) Statistical Analysis Plan Final

Template 36 Descriptive statistics of <anti-RSV A neutralizing antibody titre, anti-RSV F antibody concentration>at pre-vaccination, Day <31, 61,> <and end of 1st RSV transmission season> for pooled RSV 1D, RSV 2D and Comparator/Placebo> groups (<Adapted> PPS for immunogenicity)

| | | Each Group<br>N=XXXX |
|---------|-----------------|----------------------|
| Visit | Characteristics | Value |
| PRE | N with data | |
| | Mean | |
| | SD | |
| | Q1 | |
| | Median | |
| | Q3 | |
| | 95% CI | (xx.x; xx.x) |
| PI(D8) | | , , , |
| PI(D31) | | |
| PI(D61) | | |
| PI(D91) | *** | |

Short group label = long group label

N = total number of subjects

N with data = number of subjects with available results

Value = value of the considered parameter

SD = standard deviation

Q1 and Q3 = 1st and 3rd quantiles

LL, UL = Exact 95% Lower and Upper confidence limits

PRE= Pre-vaccination

D31 = Post-vaccination at Day 31

D61 = Post-vaccination at Day 61

Template 37 Reverse cumulative distribution curves for anti-RSV-A neutralising antibody titres in each group at baseline and <Day 31, Day 61, End of first RSV season> for pooled RSV 1D, RSV 2D and Comparator/Placebo> group <PPS for analysis of immunogenicity at <Day X, End of 1st RSV season>



Short group label = long group label

Template 38 Individual results of anti-RSV-A neutralising antibody titre at Day <61/end of first RSV season> versus pre-vaccination in <each pooled <RSV 1D, RSV 2D> group> and Comparator/placebo group> (PPS for analysis of immunogenicity at <Day X>)



Short group label = long group label

Note: This graph is provided as an example. The same graph will be generated for each assay and each timepoint separately (Days 61, end of first RSV season)

Template 39 Number and percentage of subjects with at least one RSV infection, RSV-RTI, RSV-LRTI, RSV-severe LRTI, RSV-very severe LRTI, All-cause LRTI and RSV hospitalization (based on WHO case definition) from vaccination dose 1 up to end of <first, second> RSV season for pooled RSV 1D, RSV 2D and Comparator/Placebo group (<Exposed Set, Exposed Set with a negative RSV exposure status>)

| | | <ea< th=""><th>ch gro</th><th>ıb&gt;</th><th colspan="4">Total<br/>N =</th></ea<> | ch gro | ıb> | Total<br>N = | | | |
|---|---|---|---|---|---|---|---|---|
| | | | 95 | | | 95 | % CI | |
| Categories | n | 0/ 1.1 | | | | % | LL | UL |
| No infection | | | | | | | | |
| RSV-infection symptomatic or asymptomatic* | | | | | | | | |
| RSV-RTI | | | | | | | | |
| RSV-LRTI | | | | | | | | |
| RSV-severe LRTI | | | | | | | | |
| RSV-very severe LRTI | | | | | | | | |
| All-cause LRTI | | | | | | | | |
| RSV hospitalization** | | | | | | | | |

Short group label = long group label

N = number of subjects with at least one administered dose

n/%= number/percentage of subjects reporting at least once the symptom

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

Template 40 Proportion of subjects with at least one RSV hospitalization over the number of subjects with at least one RSV infection (symptomatic or asymptomatic\*) from vaccination dose 1 up to end of <first, second> RSV season for pooled RSV 1D, RSV 2D and Comparator/Placebo group <Exposed Set, Exposed Set with negative RSV baseline status>

| | | <each group=""> N= 95 % CI</each> | | |
|---|---|---|---|---|
| | | | | 95 % CI |
| Symptom | n | % | LL | UL |
| RSV hospitalization** | | | | |

Short group label = long group label

N= number of subjects with at least one RSV infection (symptomatic or asymptomatic)

n/%= number/percentage of subjects reporting at least one RSV hospitalization

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

<sup>\*</sup> Association to RSV based on central testing only for asymptomatic visit (no local test available)

<sup>\*\*</sup> Confirmed RSV infection and hospitalized for acute medical condition

<sup>\*</sup> Association to RSV based on central testing only for asymptomatic visit (no local test available)

<sup>\*\*</sup> Confirmed RSV infection and hospitalized for acute medical condition

204894 (RSV-PED-011) Statistical Analysis Plan Final

Template 41 Number and percentage of subjects reporting the RSV infection of different severity (based on WHO case definition) by number of events experienced between vaccination dose 1 up to end of <first, second> RSV season for pooled RSV 1D, RSV 2D and Comparator/Placebo group <Exposed Set, Exposed Set with negative RSV baseline status>

| | | <each group=""><br/>N=xx</each> | | | |
|---|---|---|---|---|---|
| | | | | 95% C | |
| Characteristics | Categories | n | % | LL | UL |
| RSV infection-symptomatic or asymptomatic* | 0 | | | | |
| | 1 | | | | |
| | 2 | | | | |
| RSV-RTI | 0 | | | | |
| | 1 | | | | |
| RSV-LRTI | 0 | | | | |
| | 1 | | | | |
| | 2 | | | | |
| RSV-Severe LRTI | 0 | | | | |
| | 1 | | | | |
| RSV-very severe LRTI | 0 | | | | |
| · | 1 | | | | |
| All cause LRTI | 0 | | | | |
| | 1 | | | | |
| | 2 | | | | |
| | 3 | | | | |
| RSV hospitalization\$ | 0 | | | | |
| · | 1 | | | | |
| | 2 | | | | |
| | 3 | | | | |

Short group label = long group label

N = number of subjects in each group

n = number of subjects in a given category

<sup>% =100\*</sup>n/N

LL, UL for percentage = Exact 95% Lower and Upper confidence limits

Please note – Single episode can be considered in multiple category depending on the symptom experienced

<sup>\*</sup> Association to RSV based on central testing only for asymptomatic visit (no local test available)

<sup>\$</sup>Confirmed RSV infection and hospitalized for acute medical condition

Template 42 Number and percentage of RSV infections and associated disease severity (based on WHO case definition) and relative risk from vaccination dose 1 up to end of <first, second> RSV season for pooled RSV 1D, RSV 2D and Comparator/Placebo group <Exposed Set, Exposed Set with negative RSV baseline status>

| | | <eac< th=""><th>p&gt;</th><th colspan="3">Relative risk<br/>(RSV1D vs<br/>Comparator/Placebo)</th><th>Re<br/>(F<br/>Compa</th><th>s<br/>icebo)</th></eac<> | p> | Relative risk<br>(RSV1D vs<br>Comparator/Placebo) | | | Re<br>(F<br>Compa | s<br>icebo) | |
|---|---|---|---|---|---|---|---|---|---|
| Catagorias | - lo/ | 95<br>LL | % CI | Values | LL 95 | % CI<br>IUL | Values | 95%<br>LL | ₀ CI<br>UL |
| Categories RSV asymptomatic (Excluding RSV-RTI, LRTI, RSV-severe LRTI or RSV-very severe LRTI) | 11 / | | OL. | values | LL | OL. | values | <b>F- L</b> | OL . |
| RSV RTI (Excluding LRTI, RSV-severe or very severe LRTI) | | | | | | | | | |
| RSV LRTI (Excluding RSV-severe or very severe LRTI) | | | | | | | | | |
| RSV-severe LRTI (Excluding RSV-very severe LRTI) | | | | | | | | | |
| RSV-very severe LRTI | | | | | | | | | |

Short group label = long group label

N = number of RSV positive samples in each group

n\*\* = number of cases in each category

n/%= number/percentage of cases in each category

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

Please note – Single episode is considered in single category of highest severity based on the symptom experienced

Template 43 Number and percentage of RSV infections (based on WHO case definition) requiring hospitalization between vaccination dose 1 up to end of <first, second> RSV season for pooled RSV 1D, RSV 2D and Comparator/Placebo group <Exposed Set, Exposed Set with negative RSV baseline status>

| | | Gro<br>N | up<br>= | | Total<br>N = | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | 95 | % CI | | | 95% | % CI | |
| Categories | n** n % LL UL n** | | | | | N | % | LL | UL |
| RSV RTI*(Excluding LRTI, severe or very severe LRTI) | | | | | | | | | |
| RSV LRTI (Excluding severe or very severe LRTI) | | | | | | | | | |
| RSV-severe LRTI (Excluding very severe LRTI) | | | | | | | | | |
| RSV-very severe LRTI | | | | | | | | | |

Short group label = long group label

N = number of RSV infections in each group

n\*\* = number of cases in each category

n/%= number/percentage of subjects reporting at least once the case

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

<sup>\*</sup> Association to RSV based on central testing only for asymptomatic visit (no local test available)

204894 (RSV-PED-011) Statistical Analysis Plan Final

Template 44 Descriptive statistics of viral load calculated on all qRT-PCR confirmed RSV infection episodes with varying disease severity (based on WHO case definition) from vaccination dose 1 up to end of <first, second> RSV season for pooled RSV 1D, RSV 2D and Comparator/Placebo group <Exposed Set, Exposed Set with negative RSV baseline status>

| | | | Group<br>N= | |
|---|---|---|---|---|
| Symptoms | Parameters | Value | LL | UL |
| RSV asymptomatic* (Excluding RSV-RTI, RSV-LRTI, RSV-severe LRTI or RSV-very severe LRTI) | n | | | |
| | GM | | | |
| | 95% CI | | | |
| | SD | | | |
| | Q1 | | | |
| | Median | | | |
| | Q3 | | | |
| | Min/Max | | | |
| RSV RTI (Excluding RSV-LRTI, RSV-severe LRTI or RSV-very severe LRTI) | | | | |
| RSV LRTI (Excluding RSV-severe or RSV-very severe LRTI) | | | | |
| RSV-severe LRTI (Excluding RSV-very severe LRTI) | | | | |
| RSV-very severe LRTI | | | | |
| RSV hospitalization\$ | | | | |

Short group label = long group label

N = number of RSV infections episodes in each group

n= Number of events in each category

SD=Standard Deviation

Q1 and Q3 = 1st and 3rd quantiles

Min/Max = Minimum/Maximum

GM = Geometric mean

LL, UL for GM = Exact 95% Lower and Upper confidence limits

Total RSV viral load computed as RSV A Viral load + RSV B Viral load

Please note: each episode for a subject is considered to be independent. We may have multiple swab for one episode. We have considered the swab with maximum viral load from one episode for the table

Please note – Except for RSV hospitalization, single episode is considered in single category of highest severity based on the symptom experienced

Please check:- To check for cases where asymptomatic swab has been taken but the subject hasve symptoms of RTI or LRTI. In this case, asymptomatic is also considered as RSV RTI/LRTI and maximum viral load of all the episode should be considered.

<sup>\*</sup> Association to RSV based on central testing only for asymptomatic visit (no local test available)

<sup>\$</sup>Confirmed RSV infection and hospitalized for acute medical condition

204894 (RSV-PED-011) Statistical Analysis Plan Final

Template 45 Descriptive statistics of maximum viral load per subjects based on qRT-PCR confirmed episode with varying disease severity (based on WHO case definition) form vaccination dose 1 up to end of <first, second> RSV season for pooled RSV 1D, RSV 2D and Comparator/Placebo group <Exposed Set, Exposed Set with negative RSV baseline status>

| | | Eac | h Group<br>N= | ) |
|---|---|---|---|---|
| | | | 95 | % CI |
| Symptoms | Parameters | Value | LL | UL |
| RSV asymptomatic* (Excluding RSV-RTI, RSV-LRTI, RSV-severe LRTI or RSV-very severe LRTI) | n | | | |
| , | GM | | | |
| | 95% CI | | | |
| | SD | | | |
| | Q1 | | | |
| | Median | | | |
| | Q3 | | | |
| | Min/Max | | | |
| RSV RTI (Excluding RSV-LRTI, RSV-severe or RSV-very severe LRTI) | | | | |
| RSV LRTI (Excluding RSV-severe or RSV-very severe LRTI) | | | | |
| RSV-severe LRTI (Excluding RSV-very severe LRTI) | | | | |
| RSV-very severe LRTI | | | | |
| RSV hospitalization\$ | | | | |

Short group label = long group label

N = number of RSV positive subjects in each group

n= Number of subjects in each category

SD=Standard Deviation

Q1 and Q3 = 1st and 3rd quantiles

Min/Max = Minimum/Maximum

GM = Geometric mean

LL, UL for GM = Exact 95% Lower and Upper confidence limits

Total RSV viral load computed as RSV A Viral load + RSV B Viral load

Please note: Except of RSV hospitalization, the subject has been considered only once in one of the category based on the maximum severity of event experienced

<sup>\*</sup> Association to RSV based on central testing only for asymptomatic visit (no local test available)

<sup>\$</sup>Confirmed RSV infection and hospitalized for acute medical condition

204894 (RSV-PED-011) Statistical Analysis Plan Final

Template 46 Frequency of multiple respiratory pathogen for qRT-PCR confirmed RSV-RTI episodes from vaccination dose 1 up to end of <first, second> RSV season for pooled RSV 1D, RSV 2D and Comparator/Placebo groups <Exposed Set, Exposed Set with negative RSV baseline status>

| | | | Group<br>N = | | Total<br>N = | | | |
|---|---|---|---|---|---|---|---|---|
| | | | | 95% CI | | | 9 | 5% CI |
| Categories | n | % | LL | UL | n | % | LL | UL |
| Influenza Virus A/California/7/2009(H1N1) | | | | | | | | |
| Adenovirus | | | | | | | | |
| Human Coronavirus OC43 | | | | | | | | |
| Human Coronavirus 229E | | | | | | | | |
| Human Coronavirus NL63 | | | | | | | | |
| Human Coronavirus HKU1 | | | | | | | | |
| Enterovirus + Rhinovirus | | | | | | | | |
| Influenza Virus A | | | | | | | | |
| Influenza Virus B | | | | | | | | |
| Influenza Virus A (H1N1) | | | | | | | | |
| Influenza Virus A (H3N2) | | | | | | | | |
| Human bocavirus | | | | | | | | |
| Human metapneumovirus | | | | | | | | |
| Parainfluenza virus 1 | | | | | | | | |
| Parainfluenza virus 2 | | | | | | | | |
| Parainfluenza virus 3 | | | | | | | | |
| Parainfluenza virus 4 | | | | | | | | |

Short group label = long group label

N = number of qRT-PCR confirmed RSV-RTI infection episodes in each group

n = number of episodes in a given category

% =100\*n/N

LL, UL for percentage = Exact 95% Lower and Upper confidence limits

204894 (RSV-PED-011) Statistical Analysis Plan Final

Template 47 Frequency of multiple respiratory pathogen for confirmed LRTI episodes from vaccination dose 1 up to end of <first, second> RSV season for pooled RSV 1D, RSV 2D and Comparator/Placebo groups <Exposed Set, Exposed Set with negative RSV baseline status>

| | | G | Froup<br>N = | | Total<br>N = | | | |
|---|---|---|---|---|---|---|---|---|
| | | | 95% | 6 CI | 95% CI | | | |
| Categories | n | % | LL | UL | n | % | LL | UL |
| Respiratory syncytial virus | | | | | | | | |
| Influenza Virus A/California/7/2009(H1N1) | | | | | | | | |
| Adenovirus | | | | | | | | |
| Human Coronavirus OC43 | | | | | | | | |
| Human Coronavirus 229E | | | | | | | | |
| Human Coronavirus NL63 | | | | | | | | |
| Human Coronavirus HKU1 | | | | | | | | |
| Enterovirus + Rhinovirus | | | | | | | | |
| Influenza Virus A | | | | | | | | |
| Influenza Virus B | | | | | | | | |
| Influenza Virus A (H1N1) | | | | | | | | |
| Influenza Virus A (H3N2) | | | | | | | | |
| Human bocavirus | | | | | | | | |
| Human metapneumovirus | | | | | | | | |
| Parainfluenza virus 1 | | | | | | | | |
| Parainfluenza virus 2 | | | | | | | | |
| Parainfluenza virus 3 | | | | | | | | |
| Parainfluenza virus 4 | | | | | | | | |

Short group label = long group label

N = number of confirmed LRTI infection episodes in each group

n = number of episodes in a given category

% =100\*n/N

LL, UL for percentage = Exact 95% Lower and Upper confidence limits

Template 48 Listing of RSV-RTI cases identified according to WHO case definitions from vaccination dose 1 up to end of second RSV season <Exposed Set, Exposed Set with negative RSV baseline status>

| Gro | Su | Sex | Age at | Count | Si | Surveill | Epis | Do | Do | On | Sp | Respir | Cen | Cen | RSV | RSV | Sev | RSV | Hospita | RVP |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| up | b. | | episo | ry | te | ance | ode | se | se | set | 02 | atory | tral | tral | -RTI | - | ere | - | lization | resul |
| | No | | de(mo | | | type | nb | | nb. | day | | rate | test | test | | LRT | RSV | very | | t |
| | | | nth) | | | | | | | | | | RSV | RSV | | I | - | sev | | |
| | | | | | | | | | | | | | Α | В | | | LRT | ere | | |
| | | | | | | | | | | | | | | | | | I | LRT | | |
| | | | | | | | | | | | | | | | | | | ) | | |
| | | | | | | | | | | | | | | | Yes/ | Yes/ | Yes/ | Yes/ | Yes/No | |
| | | | | | | | | | | | | | | | No | No | No | No | | |

Short group label = long group label

204894 (RSV-PED-011) Statistical Analysis Plan Final

Template 49 Listing of RSV-RTI requiring hospitalization and type of inpatient facility required from vaccination dose 1 up to end of second RSV season <Exposed Set, Exposed Set with negative RSV baseline status>

| Gro | Sub | Sex | Age at | Coun | Classific | Total | No. of | No. of | No. of | No. of | No. of | No. of | RVP | Patho |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| up | No. | | episode | try | ation of | days | days of | days of | days | days | days | days | resu | gen |
| | | | (month) | | episode | hospitali | monitor | nasoga | oxygen | respirat | mechan | child | lt | identif |
| | | | | | per | zed | ing or | stric or | administ | ory | ical | kept in | | ied in |
| | | | | | WHO* | | nursing | intraven | ered | support | ventilati | paediat | | RVP |
| | | | | | | | | ous | | given | on | rics | | |
| | | | | | | | | fluids | | | given | intensiv | | |
| | | | | | | | | given | | | | e care | | |
| | | | | | | | | | | | | unit | | |
| | | | | | | | | | | | | | Yes/ | |
| | | | | | | | | | | | | | No | |

Short group label = long group label

Template 50 Number and percentage of subjects with highest associated severity of RSV infection (based on WHO case definition) from vaccination dose 1 up to <first, second> RSV season for pooled RSV 1D, RSV 2D and Comparator/Placebo groups <Exposed Set, Exposed Set with negative RSV baseline status>

| | | ( | | up | | Total<br>N = | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | N = | | | | | | 1 | N = | | |
| | 95% C | | | <u>% CI</u> | | | | 95% | % CI | |
| Categories | n** | n | % | L | UL | n** | n | % | LL | UL |
| No Infection | | | | | | | | | | |
| RSV asymptomatic (Excluding RSV-RTI, RSV-LRTI, RSV-severe LRTI | | | | | | | | | | |
| or RSV-very severe LRTI) | | | | | | | | | | |
| RSV RTI (Excluding RSV-LRTI, RSV-severe or very severe LRTI) | | | | | | | | | | |
| RSV LRTI (Excluding RSV-severe or very severe LRTI) | | | | | | | | | | |
| RSV-severe LRTI (Excluding RSV-very severe LRTI) | | | | | | | | | | |
| RSV-very severe LRTI | | | | | | | | | | |

Short group label = long group label

N = number of subjects in each group

n\*\* = number of cases in each category

n/%= number/percentage of subjects reporting at least once the case

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

Please note – Single episode can be considered in single category depending on the highest severity symptom experienced

<sup>\*</sup>subject will be classified per maximum severity experienced

204894 (RSV-PED-011) Statistical Analysis Plan Final

Template 51 Number and percentage of subjects reporting the RSV infection of maximum severity (based on WHO case definition) by number of events experienced between vaccination dose 1 up to end of <first, second> RSV season for pooled RSV 1D, RSV 2D and Comparator/Placebo groups <Exposed Set, Exposed Set with negative RSV baseline status >

| | | | | Tota | al | |
|---|---|---|---|---|---|---|
| | | | | | 9 | 5% CI |
| Characteristics | Categories | N | n | % | LL | UL |
| RSV asymptomatic (Excluding RSV-RTI, RSV-LRTI, RSV-severe LRTI or RSV-very severe LRTI) | 0 | | | | | |
| • , | 1 | | | | | |
| | 2 | | | | | |
| RSV-RTI (Excluding RSV-LRTI, RSV severe or very severe LRTI) | 0 | | | | | |
| , | 1 | | | | | |
| RSV-LRTI (Excluding RSV severe or very severe LRTI) | 0 | | | | | |
| | 1 | | | | | |
| RSV-Severe LRTI Excluding RSV very severe LRTI) | 0 | | | | | |
| , , | 1 | | | | | |
| RSV-very severe LRTI | 0 | | | | | |
| • | 1 | | | | | |

Short group label = long group label

Please note - Single episode will be considered in single category depending on the maximum severity experienced

N = number of subjects in each group

n = number of subjects in a given category

<sup>% =100\*</sup>n/N

LL, UL for percentage = Exact 95% Lower and Upper confidence limits

204894 (RSV-PED-011) Statistical Analysis Plan Final

Template 52 Number and percentage of subjects with <anti-RSV A antibody titre, anti-RSV F concentration> equal to or above <cut-off ><unit> and gm<t,c> for pooled RSV 1D, RSV 2D and Comparator/Placebo> groups – by RSV baseline status (<Adapted>PPS of immunogenicity at <Day X, end of 1st RSV season>)

| | | | | > | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Antibody | Time point | Cut- | | | | | | | <r< th=""><th>SV-ve</th><th>&gt;</th><th></th></r<> | SV-ve | > | |
| off | | | | | <rsv+\< th=""><th>/e&gt;</th><th></th><th></th><th></th><th></th><th></th><th></th></rsv+\<> | /e> | | | | | | |
| | | | | | | 959 | % CI | | | | 959 | % CI |
| | | | N | n | value | LL | UL | N | n | value | LL | UL |
| <antibody 1=""> <time 1="" point=""> <cut-%>=<cut-off 1=""> off 1&gt; <unit></unit></cut-off></cut-%></time></antibody> | | XXX | XXX | XX.X | xx.x | XX.X | XXX | XXX | XX.X | XX.X | XX.X | |
| | | GM <t,c></t,c> | XXX | | XX.X | XX.X | XX.X | XXX | | XX.X | XX.X | |
| | | | | | | | | | | | | XX.X |

Short group label = long group label

GMT/C = geometric mean antibody titer/concentration

N = Number of subjects with available results

n/% = number/percentage of subjects with titer/concentration equal to or above specified value

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

PRE= Pre-vaccination

D31 = Post-vaccination at Day 31

D61 = Post-vaccination at Day 61

RSV1S = End of 1st RSV transmission season

RSV+ve = Subjects are RSV positive at baseline

RSV-ve = Subject are RSV negative at baseline

204894 (RSV-PED-011) Statistical Analysis Plan Final

Template 53 Distribution of <RSV-A neutralising antibody titre, RSV-F antibody concentration> for pooled RSV 1D, RSV 2D and Comparator/Placebo> groups – by RSV baseline status(<Adapted>PPS for immunogenicity <at Day X, end of 1st RSV season>)

| | | | | | | | | <each g<="" th=""><th>roup&gt;</th><th></th><th></th><th></th></each> | roup> | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Antibody | Time point | Cut-off | | | <rsv+< th=""><th>/e&gt;</th><th></th><th></th><th><r< th=""><th>SV-ve&gt;</th><th></th><th></th></r<></th></rsv+<> | /e> | | | <r< th=""><th>SV-ve&gt;</th><th></th><th></th></r<> | SV-ve> | | |
| | | | | | | 95% | CI | | | | 95% | CI |
| | | | N | n | value | LL | UL | N | n | value | LL | UL |
| <antibody 1=""></antibody> | · <time 1="" point=""></time> | <cut-off 1<="" td=""><td>XXX</td><td>XXX</td><td>XX.X</td><td>XX.X</td><td>XX.X</td><td>XXX</td><td>XXX</td><td>XX.X</td><td>XX.X</td><td>XX.X</td></cut-off> | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | | >=cut-off 2 | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | | >=cut-off 3 | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | <time 2="" point=""></time> | <cut-off 1<="" td=""><td>XXX</td><td>XXX</td><td>XX.X</td><td>XX.X</td><td>XX.X</td><td>XXX</td><td>XXX</td><td>XX.X</td><td>XX.X</td><td>XX.X</td></cut-off> | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | | >=cut-off 2 | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | | >=cut-off 3 | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |

Short group label = long group label

N = number of subjects with available results

n/% = number/percentage of subjects with <titer, concentration> within the specified criterion

<95>% CI = <95>% confidence interval; LL = Lower Limit, UL = Upper Limit

PRE= Pre-vaccination

D31 = Post-vaccination at Day 31

D61 = Post-vaccination at Day 61

RSV1S = End of 1st RSV transmission season

RSV+ve = Subjects are RSV positive at baseline

RSV-ve = Subject are RSV negative at baseline

204894 (RSV-PED-011) Statistical Analysis Plan Final

Template 54 Number and percentage of subjects with <anti-RSV A antibody titre, anti-RSV F concentration> equal to or above <cut-off ><unit> and GMR for pooled RSV 1D, RSV 2D and Comparator/Placebo> groups – by RSV baseline status (PPS of immunogenicity at <Day X, End of 1st RSV season>)

| | | <each group=""></each> | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Antibody | Time point | | | | | | | | | | | |
| Cut-off | | | | | <rsv+< th=""><th>-ve&gt;</th><th></th><th></th><th></th><th><rsv< th=""><th>-ve&gt;</th><th></th></rsv<></th></rsv+<> | -ve> | | | | <rsv< th=""><th>-ve&gt;</th><th></th></rsv<> | -ve> | |
| | | | 95% CI | | | | | | % CI | | | |
| | | | N | n | value | LL | UL | N | n | value | LL | UL |
| <antibody 1=""></antibody> | <time 1="" point=""></time> | %>= <cut-off 1=""> <unit></unit></cut-off> | XXX | xxx | xx.x | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| YOUL'ON IP | | GMC/T | XXX | | XX.X | xx.x | XX.X | XXX | | XX.X | XX.X | XX.X |
| | | Visit comparison / baseline | | | | | | | | | | |
| | | GMR | XXX | | XX.X | XX.X | XX.X | XXX | | XX.X | XX.X | XX.X |

Short group label = long group label

GMT = geometric mean antibody titer

N = Number of subjects with available results at the two considered time points

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

PRE= Pre-vaccination

D31 = Post-vaccination at Day 31

D61 = Post-vaccination at Day 61

RSV1S = End of 1st RSV transmission season

RSV+ve = Subjects are RSV positive at baseline

RSV-ve = Subject are RSV negative at baseline

Template 55 Descriptive statistics of <anti-RSV A neutralizing antibody titre, anti-RSV F antibody concentration>at pre-vaccination, Day <31, 61,> <and end of 1st RSV transmission season> for pooled RSV 1D, RSV 2D and Comparator/Placebo> groups – by RSV baseline status (<Adapted> PPS for immunogenicity)

| | | | Group<br>XXX |
|-------|-----------------|------------------|------------------|
| | | RSV+ve<br>N=XXXX | RSV-ve<br>N=XXXX |
| Visit | Characteristics | Value | Value |
| PRE | N with data | | |
| | Mean | | |
| | SD | | |
| | Q1 | | |
| | Median | | |
| | Q3 | | |
| | 95% CI | (xx.x; xx.x) | (xx.x; xx.x) |
| D31 | | , , , | , , , |
| D61 | | | |
| RSV1S | | | |

Short group label = long group label

N = total number of subjects

N with data = number of subjects with available results

Value = value of the considered parameter

SD = standard deviation

Q1 and Q3 = 1st and 3rd quantiles

LL, UL = Exact 95% Lower and Upper confidence limits

PRE= Pre-vaccination

D31 = Post-vaccination at Day 31

D61 = Post-vaccination at Day 61

RSV1S = End of 1st RSV transmission season

RSV+ve = Subjects are RSV positive at baseline

RSV-ve = Subject are RSV negative at baseline

Template 56 Summary of subjects by unsolicited adverse event category with onset within 30 days of first and second vaccination (Exposed Set)

| | | | up 1> | <g<br>N:</g<br> | | | | |
|---|---|---|---|---|---|---|---|---|
| | | 95% CI | | | | | 959 | % CI |
| | n | % | LL | UL | n | % | LL | UL |
| At least one unsolicited adverse event | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| At least one related unsolicited adverse event | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| At least one grade 3 unsolicited adverse event | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| At least one grade 3 related unsolicited adverse event | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |
| At least one medically attended unsolicited adverse event | XXX | XX.X | XX.X | XX.X | XXX | XX.X | XX.X | XX.X |

Any adverse event = at least one adverse event experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with at least one administered vaccination

n/% = number/percentage of subjects reporting the adverse event at least once

95% CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Template 57 Number and percentage of subjects with at least one RSV-RTI progressing to RSV-LRTI, RSV-severe LRTI, RSV-very severe LRTI and RSV hospitalization from vaccination dose 1 up to end of <first, second> RSV season for pooled RSV 1D, RSV 2D and Comparator/Placebo groups <ES, Exposed Set with negative RSV exposure status>

| | | <each group=""> N =</each> | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | 90% CI | | | | | 90% CI |
| Categories | n | % | LL | UL | n | % | LL | UL |
| RSV-LRTI | | | | | | | | |
| RSV-severe LRTI | | | | | | | | |
| RSV-very severe LRTI | | | | | | | | |
| RSV hospitalization* | | | | | | | | |

<sup>&</sup>lt;Blinded = Blinded group>

N = number of subjects with at least one RSV-RTI infection

n/%= number/percentage of subjects reporting at least once the symptom

90%CI= Exact 90% confidence interval; LL = lower limit, UL = upper limit

Please note - Single episode is considered in single category of highest severity based on the symptom experienced

<sup>&</sup>lt;RSV 1D = Pooled 1D RSV>

<sup>&</sup>lt;RSV 2D = Pooled 2D RSV>

<sup>&</sup>lt;COMP PLB = Pooled comparator or placebo>

<sup>\*</sup> Confirmed RSV infection and hospitalized for acute medical condition